CLINICAL TRIAL: NCT03617185
Title: The Effect of High Intensity Interval Training and Surgical Weight Loss on Distal Symmetric Polyneuropathy Outcomes
Brief Title: Effect of Exercise and Surgical Weight Loss on Polyneuropathy
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Michigan (Other)
Collaborators: National Institute of Diabetes and Digestive and Kidney Diseases (NIDDK) (NIH)
Responsible Party: Principal Investigator, Brian Callaghan, Fovette E Dush Early Career Professor and Assistant Professor of Neurology, University of Michigan
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: HUM00143541; 1R01DK115687-01A1 (NIH)
Record Dates: First submitted 2018-07-14; First posted 2018-08-06 (Actual); Results first posted 2025-10-29 (Actual); Last update posted 2025-10-29 (Actual); Status verified 2025-10

CONDITIONS: Polyneuropathies; Obesity; Bariatric Surgery Candidate
Keywords: Metabolic syndrome; Exercise
MeSH Terms: conditions — Polyneuropathies; Obesity; Metabolic Syndrome; Motor Activity | interventions — High-Intensity Interval Training; Bariatric Surgery

STUDY DESIGN:
Intervention Model Description: Patients will be assigned to one of 4 arms, bariatric surgery/HIIT, bariatric surgery/routine exercise, no bariatric surgery/HIIT, no bariatric surgery/routine exercise.
Who Masked: Outcomes Assessor
Masking Description: The neuropathy outcomes assessors will be blinded to the exercise protocol that the patients are randomized to and the surgical status for the duration of the study.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (4):
- Bariatric Surgery/HIIT (Active Comparator): Patients who have undergone bariatric surgery will be randomized to this arm and will follow a high intensity interval training (HIIT) protocol for 24 months. Patients will complete 2 supervised HIIT sessions and 1 unsupervised HIIT session a week.
  Interventions: Other: High Intensity Interval Training (HIIT); Procedure: Bariatric surgery
- Bariatric Surgery/Routine Exercise (Active Comparator): Patients who have undergone bariatric surgery will be randomized to this arm and will follow a standard routine exercise regimen for 24 months.
  Interventions: Other: Routine Exercise; Procedure: Bariatric surgery
- No Bariatric Surgery/HIIT (Active Comparator): Patients who have not undergone bariatric surgery will be randomized to this arm and will follow a high intensity interval training (HIIT) protocol for 24 months. Patients will complete 2 supervised HIIT sessions and 1 unsupervised HIIT session a week.
  Interventions: Other: High Intensity Interval Training (HIIT)
- No Bariatric Surgery/Routine Exercise (Active Comparator): Patients who have not undergone bariatric surgery will be randomized to this arm and will follow a standard routine exercise regimen for 24 months.
  Interventions: Other: Routine Exercise

INTERVENTIONS:
Other: High Intensity Interval Training (HIIT) — Patients will complete a HIIT training protocol of a total of 10 x 1 min intervals at 90% heart rate (HR) max. They will continue this training protocol, 3 sessions a week (2 supervised and 1 unsupervised), for 24 months.
  Arms: Bariatric Surgery/HIIT; No Bariatric Surgery/HIIT
Other: Routine Exercise — Patients will receive counseling regarding exercise as a routine part of their participation in the bariatric surgery clinic. Specifically, they are counseled to participate in 60 min of aerobic exercise daily in addition to 2-3 non-consecutive days of strength training workouts every wk. Patients are encouraged to contact the bariatric conditioning program, obtain a gym membership, purchase exercise equipment, join a walking group, and/or sign up for fitness classes (employer or city parks and recreation).
  Arms: Bariatric Surgery/Routine Exercise; No Bariatric Surgery/Routine Exercise
Procedure: Bariatric surgery — Patients will undergo bariatric surgery as part of their routine care
  Arms: Bariatric Surgery/HIIT; Bariatric Surgery/Routine Exercise

SUMMARY:
The purpose of this research study is to evaluate how exercise and surgical weight loss affect how likely an individual is to develop peripheral neuropathy and other neurologic complications.

DETAILED DESCRIPTION:
The length of this study, including screening is approximately 24 months. Patients at Bariatric Surgery Clinics will be recruited for this study. Both patients that decide to undergo bariatric surgery, and those that do not undergo surgery will be enrolled. Patients will be randomized to either a high intensity interval training (HIIT) or standard exercise regimen after eligibility is confirmed and the baseline visit is complete. All patients will complete follow-up appointments at 3 month, 12 months and 24 months. Patients that are randomized to the HIIT program will compete 2 supervised and 1 unsupervised training sessions a week for 24 months.

ELIGIBILITY:
Inclusion Criteria:

* Attending a bariatric surgery clinic
* BMI > 35 with one comorbid condition present or BMI > 40 without comorbid conditions present
* Willing and capable to sign the Institutional Review Board (IRB) approved consent form and cooperate with the medical procedures for the study duration
* Willing to accept random treatment assignment to HIIT or routine exercise counseling

Exclusion Criteria:

* History of distal symmetric polyneuropathy (DSP) from causes other than diabetes and/or the metabolic syndrome as determined through medical history, family history, history of medications, occupational history, history of exposure to toxins, physical and neurological examinations;
* Use of warfarin, heparin, or other anticoagulants, which would increase the risk of complications from skin biopsy
* Contraindication to HIIT participation including a failed exercise stress test
* Participation in an experimental medication trial within 3 months of starting the study
* Undergoing therapy for malignant disease other than basal-cell or squamous-cell skin cancer
* Medical or psychiatric reason for not being a surgical candidate
* Requiring a walking assist device;
* Currently smoking

Min Age: 40 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 140 (Actual)
Dates: Start 2018-07-12 (Actual); Primary Completion 2024-08-01 (Actual); Study Completion 2024-08-01 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Brian C Callaghan, MD, MS, Principal Investigator — University of Michigan, Department of Neurology
Locations (1):
- University Of Michigan, Ann Arbor, Michigan, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Reynolds EL, Koenig F, Watanabe M, Kwiatek A, Elafros MA, Stino A, Henderson D, Herrmann DN, Feldman EL, Callaghan BC. Comparison of intraepidermal nerve fiber density and confocal corneal microscopy for neuropathy. Ann Clin Transl Neurol. 2024 Dec;11(12):3115-3124. doi: 10.1002/acn3.52218. Epub 2024 Oct 12. PMID 39394845

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Participants were recruited from Bariatric Surgery clinics in Ann Arbor and Detroit.
Pre-assignment Details: 140 participants were randomized to one of the four arms. Prior to randomization, participants had a screening visit, pre-baseline visit, and baseline visit to confirm eligibility. If participants qualified for the study, they were randomized and moved on with the study.
Groups:
- Bariatric Surgery/HIIT: High Intensity Interval Training (HIIT) Patients will complete a HIIT training protocol of a total of 10 x 1 min intervals at 90% heart rate (HR) max. They will continue this training protocol, 3 sessions a week (2 supervised and 1 unsupervised), for 24 months.
  Procedure/Surgery: Bariatric surgery Patients will undergo bariatric surgery as part of their routine care.
- No Bariatric Surgery/HIIT: High Intensity Interval Training (HIIT) Patients will complete a HIIT training protocol of a total of 10 x 1 min intervals at 90% heart rate (HR) max. They will continue this training protocol, 3 sessions a week (2 supervised and 1 unsupervised), for 24 months.
  Procedure/Surgery: None
- Bariatric Surgery/Routine Exercise: Routine Exercise Patients will receive counseling regarding exercise as a routine part of their participation in the bariatric surgery clinic. Specifically, they are counseled to participate in 60 min of aerobic exercise daily in addition to 2-3 non-consecutive days of strength training workouts every wk. Patients are encouraged to contact the bariatric conditioning program, obtain a gym membership, purchase exercise equipment, join a walking group, and/or sign up for fitness classes (employer or city parks and recreation).
  Procedure/Surgery: Bariatric surgery Patients will undergo bariatric surgery as part of their routine care.
- No Bariatric Surgery/Routine Exercise: Routine Exercise Patients will receive counseling regarding exercise as a routine part of their participation in the bariatric surgery clinic. Specifically, they are counseled to participate in 60 min of aerobic exercise daily in addition to 2-3 non-consecutive days of strength training workouts every wk. Patients are encouraged to contact the bariatric conditioning program, obtain a gym membership, purchase exercise equipment, join a walking group, and/or sign up for fitness classes (employer or city parks and recreation).
  Procedure/Surgery: None
Period: Baseline
Arm/Group | Bariatric Surgery/HIIT | No Bariatric Surgery/HIIT | Bariatric Surgery/Routine Exercise | No Bariatric Surgery/Routine Exercise
Started | 35 | 35 | 35 | 35
Completed | 35 | 32 | 32 | 32
Not Completed | 0 | 3 | 3 | 3
Not completed — Lost to Follow-up | 0 | 2 | 1 | 1
Not completed — Withdrawal by Subject | 0 | 1 | 0 | 1
Not completed — Driving Distance/Travel | 0 | 0 | 2 | 0
Not completed — Family Obligations | 0 | 0 | 0 | 1
Period: 3 Months
Arm/Group | Bariatric Surgery/HIIT | No Bariatric Surgery/HIIT | Bariatric Surgery/Routine Exercise | No Bariatric Surgery/Routine Exercise
Started | 35 | 32 | 32 | 32
Completed | 29 | 28 | 32 | 29
Not Completed | 6 | 4 | 0 | 3
Not completed — Lost to Follow-up | 4 | 1 | 0 | 2
Not completed — Withdrawal by Subject | 1 | 3 | 0 | 0
Not completed — Driving Distance/Travel | 1 | 0 | 0 | 0
Not completed — Family Obligations | 0 | 0 | 0 | 1
Period: 12 Months
Arm/Group | Bariatric Surgery/HIIT | No Bariatric Surgery/HIIT | Bariatric Surgery/Routine Exercise | No Bariatric Surgery/Routine Exercise
Started | 29 | 28 | 32 | 29
Completed | 26 | 27 | 28 | 28
Not Completed | 3 | 1 | 4 | 1
Not completed — Lost to Follow-up | 3 | 1 | 3 | 0
Not completed — Withdrawal by Subject | 0 | 0 | 0 | 1
Not completed — Driving Distance/Travel | 0 | 0 | 1 | 0
Period: 24 Months
Arm/Group | Bariatric Surgery/HIIT | No Bariatric Surgery/HIIT | Bariatric Surgery/Routine Exercise | No Bariatric Surgery/Routine Exercise
Started | 26 | 27 | 28 | 28
Completed (Anyone who did not complete visit 6 was considered withdrawn after visit 5.) | 26 | 27 | 28 | 28
Not Completed | 0 | 0 | 0 | 0

BASELINE CHARACTERISTICS:
Population: Data was collected for participants who were randomized in the study
Groups:
- Total: Total of all reporting groups
Arm/Group | No Bariatric Surgery/HIIT | Bariatric Surgery/Routine Exercise | Bariatric Surgery/HIIT | No Bariatric Surgery/Routine Exercise | Total
Number analyzed (Participants) | 35 | 35 | 35 | 35 | 140
Age, Continuous [Median (Standard Deviation); unit: years] | 50.54 (7.56) | 49.66 (6.98) | 49.91 (5.77) | 51.14 (8.08) | 50.31 (7.1)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 29 | 26 | 28 | 25 | 108
  Male | 6 | 9 | 7 | 10 | 32
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 2 | 0 | 0 | 1 | 3
  Not Hispanic or Latino | 33 | 35 | 35 | 34 | 137
  Unknown or Not Reported | 0 | 0 | 0 | 0 | 0
Race/Ethnicity, Customized [Count of Participants; unit: Participants]
  Asian | 0 | 0 | 0 | 1 | 1
  Bi/Multi Racial Non-Hispanic | 0 | 0 | 1 | 0 | 1
  Black | 13 | 2 | 5 | 14 | 34
  Hispanic | 1 | 0 | 0 | 1 | 2
  Hispanic White | 1 | 0 | 0 | 0 | 1
  Middle Eastern | 0 | 0 | 0 | 1 | 1
  Native-American | 0 | 0 | 0 | 1 | 1
  Native-American/Black | 1 | 1 | 0 | 0 | 2
  Non-Hispanic White | 19 | 32 | 29 | 17 | 97

OUTCOME MEASURES:

1. Primary Outcome: Intraepidermal Nerve Fiber Density (IENFD) at the Proximal Thigh
Description: Intraepidermal Nerve Fiber Density (IENFD) as assessed by 3mm skin biopsies at the proximal thigh.
Time Frame: Baseline, 3 months, 12 months and 24 months
Population: The number analyzed the number of participants that completed the outcome at each respective visit. This number will not include participants dropped out, missed a visit, or declined the particular outcome measure.
Measure: Mean (Standard Deviation); unit: fibers/mm
Arm/Group | Bariatric Surgery/HIIT | Bariatric Surgery/Routine Exercise | No Bariatric Surgery/HIIT | No Bariatric Surgery/Routine Exercise
Number analyzed (Participants) | 35 | 35 | 35 | 35
fibers/mm
  Baseline | 11.9 (3.9) | 12.7 (4.4) | 9.8 (4.9) | 11 (4.6)
  3 Months: number analyzed (Participants) | 35 | 32 | 32 | 32
  3 Months | 12.6 (3.9) | 14.3 (5) | 9.9 (4.2) | 10.6 (6)
  12 Months: number analyzed (Participants) | 29 | 32 | 28 | 29
  12 Months | 11.5 (6.1) | 14.2 (6.2) | 9.2 (4.2) | 8.5 (4.4)
  24 Months: number analyzed (Participants) | 26 | 28 | 27 | 28
  24 Months | 11.9 (6.0) | 13.5 (6.2) | 10.3 (4.3) | 9.3 (3.8)
Statistical Analysis 1: Comparison: Bariatric Surgery/HIIT vs No Bariatric Surgery/Routine Exercise; Test type: Superiority; p = 0.15, t-test, 2 sided — The P-value tests whether the within-participant change in the outcome from baseline to 2 years differs between the treatment and no-treatment groups; Mean Difference (Net) = -1.98, 95% CI 2-sided [-4.63 to 0.74]
Statistical Analysis 2: Comparison: Bariatric Surgery/Routine Exercise vs No Bariatric Surgery/Routine Exercise; Test type: Superiority; p = 0.08, t-test, 2 sided — [p-value comment as in outcome 1, analysis 1]; Mean Difference (Net) = -2.33, 95% CI 2-sided [-4.98 to 0.31]
Statistical Analysis 3: Comparison: No Bariatric Surgery/HIIT vs No Bariatric Surgery/Routine Exercise; Test type: Superiority; p = 0.15, t-test, 2 sided — [p-value comment as in outcome 1, analysis 1]; Mean Difference (Net) = -1.84, 95% CI 2-sided [-4.43 to 0.74]
Statistical Analysis 4: Comparison: Bariatric Surgery/HIIT vs No Bariatric Surgery/Routine Exercise; Test type: Superiority; p = 0.67, Mixed Models Analysis — The P-value tests for association between the outcome and treatment at each visit, compared to the no-treatment group; Interaction term for difference in slope = 0.07, 95% CI 2-sided [-0.02 to 0.16]
Statistical Analysis 5: Comparison: Bariatric Surgery/Routine Exercise vs No Bariatric Surgery/Routine Exercise; Test type: Superiority; p = 0.77, Mixed Models Analysis — The P-value tests for association between the outcome and treatment at each visit, compared to the no-treatment group; Interaction term for difference in slope = 0.09, 95% CI 2-sided [0.002 to 0.19]
Statistical Analysis 6: Comparison: No Bariatric Surgery/HIIT vs No Bariatric Surgery/Routine Exercise; Test type: Superiority; p = 0.69, Mixed Models Analysis — The P-value tests for association between the outcome and treatment at each visit, compared to the no-treatment group; Interaction term for difference in slope = 0.07, 95% CI 2-sided [-0.02 to 0.16]

2. Secondary Outcome: Intraepidermal Nerve Fiber Density (IENFD) at Distal Leg.
Description: Intraepidermal Nerve Fiber Density (IENFD) as assessed by 3mm skin biopsies at the distal leg.
Time Frame: Baseline, 3 months, 12 months and 24 months
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: fibers/mm
Arm/Group | Bariatric Surgery/HIIT | Bariatric Surgery/Routine Exercise | No Bariatric Surgery/HIIT | No Bariatric Surgery/Routine Exercise
Number analyzed (Participants) | 35 | 35 | 35 | 35
fibers/mm
  Baseline | 6.3 (4) | 6.8 (4.3) | 7.3 (4.1) | 5.7 (3.8)
  3 Months: number analyzed (Participants) | 35 | 32 | 32 | 32
  3 Months | 7.3 (4.1) | 6.2 (4.1) | 6.3 (3.6) | 5.5 (3.8)
  12 Months: number analyzed (Participants) | 29 | 32 | 28 | 29
  12 Months | 7.7 (5.2) | 8.7 (5.4) | 6.4 (3.6) | 6.4 (5.5)
  24 Months: number analyzed (Participants) | 26 | 28 | 27 | 28
  24 Months | 6.9 (4.5) | 7.4 (4.4) | 6.4 (3.8) | 5.8 (4.1)
Statistical Analysis 1: Comparison: Bariatric Surgery/HIIT vs No Bariatric Surgery/Routine Exercise; Test type: Superiority; p = 0.27, t-test, 2 sided — [p-value comment as in outcome 1, analysis 1]; Mean Difference (Net) = -0.98, 95% CI 2-sided [-2.77 to 0.79]
Statistical Analysis 2: Comparison: Bariatric Surgery/Routine Exercise vs No Bariatric Surgery/Routine Exercise; Test type: Superiority; p = 0.18, t-test, 2 sided — [p-value comment as in outcome 1, analysis 1]; Mean Difference (Net) = -1.09, 95% CI 2-sided [-2.71 to 0.53]
Statistical Analysis 3: Comparison: No Bariatric Surgery/HIIT vs No Bariatric Surgery/Routine Exercise; Test type: Superiority; p = 0.21, t-test, 2 sided — [p-value comment as in outcome 1, analysis 1]; Mean Difference (Net) = 1.32, 95% CI 2-sided [-0.82 to 3.48]
Statistical Analysis 4: Comparison: Bariatric Surgery/HIIT vs No Bariatric Surgery/Routine Exercise; Test type: Superiority; p = 0.66, Mixed Models Analysis — The P-value tests for association between the outcome and treatment at each visit, compared to the no-treatment group; Interaction term for difference in slope = 0.02, 95% CI 2-sided [-0.05 to 0.09]
Statistical Analysis 5: Comparison: Bariatric Surgery/Routine Exercise vs No Bariatric Surgery/Routine Exercise; Test type: Superiority; p = 0.25, Mixed Models Analysis — The P-value tests for association between the outcome and treatment at each visit, compared to the no-treatment group; Interaction term for difference in slope = 0.05, 95% CI 2-sided [-0.02 to 0.11]
Statistical Analysis 6: Comparison: No Bariatric Surgery/HIIT vs No Bariatric Surgery/Routine Exercise; Test type: Superiority; p = 0.09, Mixed Models Analysis — The P-value tests for association between the outcome and treatment at each visit, compared to the no-treatment group; Interaction term for difference in slope = -0.06, 95% CI 2-sided [-0.13 to 0.01]

3. Secondary Outcome: Corneal Confocal Microscopy (CCM) - Fiber Density
Description: Non-invasive imaging technique of the corneal nerves to quantify nerve density and morphology.
  Corneal Nerve Fiber Density are quantified by fibers/mm2, a higher number represents a higher density of fibers. Lower numbers indicate worse neuropathy.
Time Frame: Baseline, 3 month, 12 months and 24 months
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: fibers/mm^2
Arm/Group | Bariatric Surgery/HIIT | Bariatric Surgery/Routine Exercise | No Bariatric Surgery/HIIT | No Bariatric Surgery/Routine Exercise
Number analyzed (Participants) | 35 | 35 | 35 | 35
fibers/mm^2
  Baseline-Corneal Nerve Fiber Density (fibers/mm2) | 22.1 (6.8) | 19.5 (5.7) | 19.5 (6.2) | 22.4 (5.4)
  3 Months-Corneal Nerve Fiber Density (fibers/mm2): number analyzed (Participants) | 35 | 32 | 32 | 32
  3 Months-Corneal Nerve Fiber Density (fibers/mm2) | 20 (6.5) | 19.9 (4.9) | 19.3 (6.5) | 19.8 (6.3)
  12 Months-Corneal Nerve Fiber Density (fibers/mm2): number analyzed (Participants) | 29 | 32 | 28 | 29
  12 Months-Corneal Nerve Fiber Density (fibers/mm2) | 19.8 (9.4) | 20.7 (5.2) | 17.2 (6.3) | 18.8 (6.8)
  24 Months-Corneal Nerve Fiber Density (fibers/mm2): number analyzed (Participants) | 26 | 28 | 27 | 28
  24 Months-Corneal Nerve Fiber Density (fibers/mm2) | 20.5 (5.1) | 20.2 (3.9) | 19 (5.5) | 18.8 (5.7)
Statistical Analysis 1: Comparison: Bariatric Surgery/HIIT vs No Bariatric Surgery/Routine Exercise; Test type: Superiority; p = 0.97, t-test, 2 sided — [p-value comment as in outcome 1, analysis 1]; Mean Difference (Net) = 0.06, 95% CI 2-sided [-3.72 to 3.85]
Statistical Analysis 2: Comparison: Bariatric Surgery/Routine Exercise vs No Bariatric Surgery/Routine Exercise; Test type: Superiority; p = 0.03, t-test, 2 sided — [p-value comment as in outcome 1, analysis 1]; Mean Difference (Net) = -3.82, 95% CI 2-sided [-7.32 to -0.31]
Statistical Analysis 3: Comparison: No Bariatric Surgery/HIIT vs No Bariatric Surgery/Routine Exercise; Test type: Superiority; p = 0.38, t-test, 2 sided — [p-value comment as in outcome 1, analysis 1]; Mean Difference (Net) = -1.56, 95% CI 2-sided [-5.18 to 2.05]

4. Secondary Outcome: Corneal Confocal Microscopy (CCM) - Branch Density
Description: Non-invasive imaging technique of the corneal nerves to quantify nerve density and morphology.
  Corneal Nerve Branch Density are quantified by branches/mm2, a higher number represents a higher density of branches. Lower numbers indicate worse neuropathy.
Time Frame: Baseline, 3 month, 12 months and 24 months
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: branches/mm^2
Arm/Group | Bariatric Surgery/HIIT | Bariatric Surgery/Routine Exercise | No Bariatric Surgery/HIIT | No Bariatric Surgery/Routine Exercise
Number analyzed (Participants) | 35 | 35 | 35 | 35
branches/mm^2
  Baseline-Corneal Nerve Branch Density (branches/mm2) | 56.4 (30.7) | 57.1 (24.6) | 53.6 (31.9) | 54.7 (25.3)
  3 Months-Corneal Nerve Branch Density (branches/mm2): number analyzed (Participants) | 35 | 32 | 32 | 32
  3 Months-Corneal Nerve Branch Density (branches/mm2) | 62.2 (32) | 72.6 (34) | 62 (31.3) | 63.9 (37.2)
  12 Months-Corneal Nerve Branch Density (branches/mm2): number analyzed (Participants) | 29 | 32 | 28 | 29
  12 Months-Corneal Nerve Branch Density (branches/mm2) | 126.6 (68.6) | 137.4 (55.) | 101.2 (57.9) | 116.8 (79)
  24 Months-Corneal Nerve Branch Density (branches/mm2): number analyzed (Participants) | 26 | 28 | 27 | 28
  24 Months-Corneal Nerve Branch Density (branches/mm2) | 124.7 (54.3) | 129.8 (39.7) | 116.6 (49.1) | 127.1 (55.9)
Statistical Analysis 1: Comparison: Bariatric Surgery/HIIT vs No Bariatric Surgery/Routine Exercise; Test type: Superiority; p = 0.62, t-test, 2 sided — [p-value comment as in outcome 1, analysis 1]
Statistical Analysis 2: Comparison: Bariatric Surgery/Routine Exercise vs No Bariatric Surgery/Routine Exercise; Test type: Superiority; p = 0.95, t-test, 2 sided — [p-value comment as in outcome 1, analysis 1]
Statistical Analysis 3: Comparison: No Bariatric Surgery/HIIT vs No Bariatric Surgery/Routine Exercise; Test type: Superiority; p = 0.59, t-test, 2 sided — [p-value comment as in outcome 1, analysis 1]

5. Secondary Outcome: Corneal Confocal Microscopy (CCM) - Fiber Length
Description: Non-invasive imaging technique of the corneal nerves to quantify nerve density and morphology.
  Corneal Nerve Fiber Length are quantified by mm/mm2, a higher number represents a higher total length of fibers. Lower numbers indicate worse neuropathy .
Time Frame: Baseline, 3 month, 12 months and 24 months
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: mm/mm2
Arm/Group | Bariatric Surgery/HIIT | Bariatric Surgery/Routine Exercise | No Bariatric Surgery/HIIT | No Bariatric Surgery/Routine Exercise
Number analyzed (Participants) | 35 | 35 | 35 | 35
mm/mm2
  Baseline-Corneal Nerve Fiber Length (mm/mm2) | 18.6 (6.1) | 18.9 (5.3) | 17.9 (6.1) | 19.3 (4.9)
  3 Months-Corneal Nerve Fiber Length (mm/mm2): number analyzed (Participants) | 35 | 32 | 32 | 32
  3 Months-Corneal Nerve Fiber Length (mm/mm2) | 19 (5.9) | 20.6 (5.3) | 19.3 (5.5) | 19.3 (6.1)
  12 Months-Corneal Nerve Fiber Length (mm/mm2): number analyzed (Participants) | 29 | 32 | 28 | 29
  12 Months-Corneal Nerve Fiber Length (mm/mm2) | 25.7 (7.5) | 28 (6.7) | 23 (8.1) | 24.7 (8.7)
  24 Months-Corneal Nerve Fiber Length (mm/mm2): number analyzed (Participants) | 26 | 28 | 27 | 28
  24 Months-Corneal Nerve Fiber Length (mm/mm2) | 25.2 (6.8) | 25.3 (4.8) | 24 (6.9) | 25.2 (7.4)
Statistical Analysis 1: Comparison: Bariatric Surgery/HIIT vs No Bariatric Surgery/Routine Exercise; Test type: Superiority; p = 0.89, t-test, 2 sided — [p-value comment as in outcome 1, analysis 1]; Mean Difference (Net) = 0.3, 95% CI 2-sided [-4.26 to 4.86]
Statistical Analysis 2: Comparison: Bariatric Surgery/Routine Exercise vs No Bariatric Surgery/Routine Exercise; Test type: Superiority; p = 0.83, t-test, 2 sided — [p-value comment as in outcome 1, analysis 1]; Mean Difference (Net) = -0.43, 95% CI 2-sided [-4.64 to 3.76]
Statistical Analysis 3: Comparison: No Bariatric Surgery/HIIT vs No Bariatric Surgery/Routine Exercise; Test type: Superiority; p = 0.82, t-test, 2 sided — [p-value comment as in outcome 1, analysis 1]; Mean Difference (Net) = 0.51, 95% CI 2-sided [-4.27 to 5.3]
Statistical Analysis 4: Comparison: Bariatric Surgery/HIIT vs No Bariatric Surgery/Routine Exercise; Test type: Superiority; p = 0.51, Mixed Models Analysis — The P-value tests for association between the outcome and treatment at each visit, compared to the no-treatment group; Interaction term for difference in slope = 0.05, 95% CI 2-sided [-0.11 to 0.21]
Statistical Analysis 5: Comparison: Bariatric Surgery/Routine Exercise vs No Bariatric Surgery/Routine Exercise; Test type: Superiority; p = 0.60, Mixed Models Analysis — The P-value tests for association between the outcome and treatment at each visit, compared to the no-treatment group; Interaction term for difference in slope = 0.04, 95% CI 2-sided [-0.11 to 0.19]
Statistical Analysis 6: Comparison: No Bariatric Surgery/HIIT vs No Bariatric Surgery/Routine Exercise; Test type: Superiority; p = 0.99, Mixed Models Analysis — The P-value tests for association between the outcome and treatment at each visit, compared to the no-treatment group; Mean Difference (Net) = 0.002, 95% CI 2-sided [-0.17 to 0.17]

6. Secondary Outcome: Corneal Confocal Microscopy (CCM) - Tortuosity Coefficient
Description: Non-invasive imaging technique of the corneal nerves to quantify nerve density and morphology.
  Tortuosity Coefficient represents the total tortuosity (twisting/bending of nerves). As a coefficient the value is unitless, a higher value represents greater tortuosity. Lower numbers indicate worse neuropathy.
Time Frame: Baseline, 3 month, 12 months and 24 months
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: Coefficient
Arm/Group | Bariatric Surgery/HIIT | Bariatric Surgery/Routine Exercise | No Bariatric Surgery/HIIT | No Bariatric Surgery/Routine Exercise
Number analyzed (Participants) | 35 | 35 | 35 | 35
Coefficient
  Baseline-Corneal Tortuosity (coefficient value) | 19.4 (5.6) | 19 (6.3) | 18.6 (6.7) | 19.2 (4.9)
  3 Months-Corneal Tortuosity (coefficient value): number analyzed (Participants) | 35 | 32 | 32 | 32
  3 Months-Corneal Tortuosity (coefficient value) | 17.8 (4.3) | 19.9 (5.6) | 17.7 (4.6) | 18.5 (4.9)
  12 Months-Corneal Tortuosity (coefficient value): number analyzed (Participants) | 29 | 32 | 28 | 29
  12 Months-Corneal Tortuosity (coefficient value) | 20.8 (7.2) | 20.6 (5.6) | 20.1 (7.3) | 21.4 (5.8)
  24 Months-Corneal Tortuosity (coefficient value): number analyzed (Participants) | 26 | 28 | 27 | 28
  24 Months-Corneal Tortuosity (coefficient value) | 20 (10.1) | 22 (7.8) | 21 (4.9) | 20.1 (5.6)
Statistical Analysis 1: Comparison: Bariatric Surgery/HIIT vs No Bariatric Surgery/Routine Exercise; Test type: Superiority; p = 0.82, t-test, 2 sided — [p-value comment as in outcome 1, analysis 1]
Statistical Analysis 2: Comparison: Bariatric Surgery/Routine Exercise vs No Bariatric Surgery/Routine Exercise; Test type: Superiority; p = 0.21, t-test, 2 sided — [p-value comment as in outcome 1, analysis 1]
Statistical Analysis 3: Comparison: No Bariatric Surgery/HIIT vs No Bariatric Surgery/Routine Exercise; Test type: Superiority; p = 0.33, t-test, 2 sided — [p-value comment as in outcome 1, analysis 1]

7. Secondary Outcome: 24-2 Frequency Doubling Technology (FDT) - Mean Deviation
Description: 24-2 FDT was used to evaluate retinopathy using visual field deficits. Mean Deviation is presented below.
  Mean deviation is the average difference from normal expected value in the patients' particular age group. Lower values indicate more visual deficit. Higher values indicate fewer visual deficit.
Time Frame: Baseline, 3 month, 12 months and 24 months
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: dB
Arm/Group | Bariatric Surgery/HIIT | Bariatric Surgery/Routine Exercise | No Bariatric Surgery/HIIT | No Bariatric Surgery/Routine Exercise
Number analyzed (Participants) | 35 | 35 | 35 | 35
dB
  Baseline-Mean Deviation | -1.6 (4.2) | -1.6 (2.7) | -2 (4.1) | -2.5 (4)
  3 Months-Mean Deviation: number analyzed (Participants) | 35 | 32 | 32 | 32
  3 Months-Mean Deviation | -1 (4.1) | -1.5 (2.7) | -1.7 (4) | -2.8 (4.6)
  12 Months-Mean Deviation: number analyzed (Participants) | 29 | 32 | 28 | 29
  12 Months-Mean Deviation | -0.9 (3.2) | -1.3 (3.1) | -2.4 (3.8) | -1.5 (4.3)
  24 Months-Mean Deviation: number analyzed (Participants) | 26 | 28 | 27 | 28
  24 Months-Mean Deviation | -1.1 (3.8) | -0.7 (2.7) | -2.3 (3.4) | -2.1 (4.8)
Statistical Analysis 1: Comparison: Bariatric Surgery/HIIT vs No Bariatric Surgery/Routine Exercise; Test type: Superiority; p = 0.98, t-test, 2 sided — [p-value comment as in outcome 1, analysis 1]; Mean Difference (Net) = 0.02, 95% CI 2-sided [-2.12 to 2.17]
Statistical Analysis 2: Comparison: Bariatric Surgery/Routine Exercise vs No Bariatric Surgery/Routine Exercise; Test type: Superiority; p = 0.71, t-test, 2 sided — [p-value comment as in outcome 1, analysis 1]; Mean Difference (Net) = -0.35, 95% CI 2-sided [-2.26 to 1.56]
Statistical Analysis 3: Comparison: No Bariatric Surgery/HIIT vs No Bariatric Surgery/Routine Exercise; Test type: Superiority; p = 0.92, t-test, 2 sided — [p-value comment as in outcome 1, analysis 1]; Mean Difference (Net) = 0.10, 95% CI 2-sided [-2.10 to 2.31]
Statistical Analysis 4: Comparison: Bariatric Surgery/HIIT vs No Bariatric Surgery/Routine Exercise; Test type: Superiority; p = 0.98, Mixed Models Analysis — The P-value tests for association between the outcome and treatment at each visit, compared to the no-treatment group; Interaction term for difference of slope = 0.001, 95% CI 2-sided [-0.08 to 0.08]
Statistical Analysis 5: Comparison: Bariatric Surgery/Routine Exercise vs No Bariatric Surgery/Routine Exercise; Test type: Superiority; p = 0.66, Mixed Models Analysis — The P-value tests for association between the outcome and treatment at each visit, compared to the no-treatment group; Interaction term for difference in slope = 0.02, 95% CI 2-sided [-0.06 to 0.10]
Statistical Analysis 6: Comparison: No Bariatric Surgery/HIIT vs No Bariatric Surgery/Routine Exercise; Test type: Superiority; p = 0.66, Mixed Models Analysis — The P-value tests for association between the outcome and treatment at each visit, compared to the no-treatment group; Interaction term for difference in slope = -0.02, 95% CI 2-sided [-0.10 to 0.06]

8. Secondary Outcome: 24-2 Frequency Doubling Technology (FDT) - Foveal Sensitivity dB
Description: 24-2 FDT was used to evaluate retinopathy using visual field deficits. Foveal sensitivity is presented below.
  Foveal sensitivity is the measurement of the fovea's light detection ability. Lower values suggest visual field deficits.
Time Frame: Baseline, 3 month, 12 months and 24 months
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: dB
Arm/Group | Bariatric Surgery/HIIT | Bariatric Surgery/Routine Exercise | No Bariatric Surgery/HIIT | No Bariatric Surgery/Routine Exercise
Number analyzed (Participants) | 35 | 35 | 35 | 35
dB
  Baseline-Foveal Sensitivity | 27.7 (4.5) | 28.3 (3.5) | 26.9 (4.9) | 25.4 (5.9)
  3 Months--Foveal Sensitivity: number analyzed (Participants) | 35 | 32 | 32 | 32
  3 Months--Foveal Sensitivity | 28.3 (5.3) | 28.3 (4.5) | 27.1 (4.1) | 26.4 (4.6)
  12 Months--Foveal Sensitivity: number analyzed (Participants) | 29 | 32 | 28 | 29
  12 Months--Foveal Sensitivity | 28.1 (4) | 28.9 (3.6) | 25.9 (5.5) | 28.3 (4.6)
  24 Months--Foveal Sensitivity: number analyzed (Participants) | 26 | 28 | 27 | 28
  24 Months--Foveal Sensitivity | 27 (5.3) | 28.2 (4.5) | 26.7 (5) | 26.5 (6.6)
Statistical Analysis 1: Comparison: Bariatric Surgery/HIIT vs No Bariatric Surgery/Routine Exercise; Test type: Superiority; p = 0.26, t-test, 2 sided — [p-value comment as in outcome 1, analysis 1]
Statistical Analysis 2: Comparison: Bariatric Surgery/Routine Exercise vs No Bariatric Surgery/Routine Exercise; Test type: Superiority; p = 0.58, t-test, 2 sided — [p-value comment as in outcome 1, analysis 1]
Statistical Analysis 3: Comparison: No Bariatric Surgery/HIIT vs No Bariatric Surgery/Routine Exercise; Test type: Superiority; p = 0.97, t-test, 2 sided — [p-value comment as in outcome 1, analysis 1]

9. Secondary Outcome: 24-2 Frequency Doubling Technology (FDT) - Pattern SD
Description: 24-2 FDT was used to evaluate retinopathy using visual field deficits. Pattern SD (PSD) is presented below.
  PSD provides information about localized loss. A higher PSD indicates a non-uniform sensitivity loss and visual field deficit.
Time Frame: Baseline, 3 month, 12 months and 24 months
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: dB
Arm/Group | Bariatric Surgery/HIIT | Bariatric Surgery/Routine Exercise | No Bariatric Surgery/HIIT | No Bariatric Surgery/Routine Exercise
Number analyzed (Participants) | 35 | 35 | 35 | 35
dB
  Baseline-Patter SD | 3.4 (1.1) | 3.1 (1.1) | 3.3 (1.1) | 3.7 (1.3)
  3 Months-Patter SD: number analyzed (Participants) | 35 | 32 | 32 | 32
  3 Months-Patter SD | 3.1 (1.1) | 3.2 (1.3) | 3.3 (1) | 3.9 (1.7)
  12 Months-Patter SD: number analyzed (Participants) | 29 | 32 | 28 | 29
  12 Months-Patter SD | 3.2 (1.1) | 3.3 (1.7) | 3.5 (1.1) | 3.6 (1.6)
  24 Months-Patter SD: number analyzed (Participants) | 26 | 28 | 27 | 28
  24 Months-Patter SD | 3.2 (0.8) | 3.1 (0.7) | 3.5 (1.1) | 3.9 (1.7)
Statistical Analysis 1: Comparison: Bariatric Surgery/HIIT vs No Bariatric Surgery/Routine Exercise; Test type: Superiority; p = 0.25, t-test, 2 sided — [p-value comment as in outcome 1, analysis 1]
Statistical Analysis 2: Comparison: Bariatric Surgery/Routine Exercise vs No Bariatric Surgery/Routine Exercise; Test type: Superiority; p = 0.98, t-test, 2 sided — [p-value comment as in outcome 1, analysis 1]
Statistical Analysis 3: Comparison: No Bariatric Surgery/HIIT vs No Bariatric Surgery/Routine Exercise; Test type: Superiority; p = 0.88, t-test, 2 sided — [p-value comment as in outcome 1, analysis 1]

10. Secondary Outcome: Retinal Fundus Photography
Description: As assessed by fundus photographs, participants were identified as either having retinopathy or not having retinopathy. Data is shown as number of people with retinopathy at a particular study visit.
Time Frame: Baseline, 3 month, 12 months and 24 months
Population: as for outcome 1
Measure: Count of Participants; unit: Participants
Arm/Group | Bariatric Surgery/HIIT | Bariatric Surgery/Routine Exercise | No Bariatric Surgery/HIIT | No Bariatric Surgery/Routine Exercise
Number analyzed (Participants) | 35 | 35 | 35 | 35
Participants
  Baseline | 0 | 1 | 1 | 1
  3 Months: number analyzed (Participants) | 35 | 32 | 32 | 32
  3 Months | 0 | 0 | 0 | 0
  12 Months: number analyzed (Participants) | 29 | 32 | 28 | 29
  12 Months | 0 | 0 | 0 | 0
  24 Months: number analyzed (Participants) | 26 | 28 | 27 | 28
  24 Months | 0 | 0 | 0 | 0
Statistical Analysis 1: Comparison: Bariatric Surgery/HIIT vs No Bariatric Surgery/Routine Exercise; Test type: Superiority; p = 1, Fisher Exact — The P-value tests whether the change in participant count (as either having retinopathy or not having retinopathy) from baseline to 2 years differs between the treatment and no-treatment groups
Statistical Analysis 2: Comparison: Bariatric Surgery/Routine Exercise vs No Bariatric Surgery/Routine Exercise; Test type: Superiority; p = 1, Fisher Exact — [p-value comment as in outcome 10, analysis 1]
Statistical Analysis 3: Comparison: No Bariatric Surgery/HIIT vs No Bariatric Surgery/Routine Exercise; Test type: Superiority; p = 0.44, Fisher Exact — [p-value comment as in outcome 10, analysis 1]

11. Secondary Outcome: Nerve Conduction Study (NCS) - Latency
Description: Latency measures the time in millisecond between stimulation and the recording electrode. Was performed on sural, peroneal, and tibial nerves. No response and abnormal values indicate neuropathy.
  * Peroneal: 0 - No response, >6.5 - Abnormal
  * Sural: 0 - No response, >4.5 - Abnormal
  * Tibial: 0 - No response, >6.1 - Abnormal
Time Frame: Baseline and 24 months
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: ms
Arm/Group | Bariatric Surgery/HIIT | Bariatric Surgery/Routine Exercise | No Bariatric Surgery/HIIT | No Bariatric Surgery/Routine Exercise
Number analyzed (Participants) | 35 | 35 | 35 | 35
ms
  Baseline-Peroneal distal motor latency (ms) | 4.6 (0.8) | 4.4 (0.6) | 4.4 (0.7) | 4.5 (1)
  Baseline-Sural peak latency (ms) | 3.8 (0.5) | 3.7 (0.4) | 3.6 (0.3) | 3.9 (0.4)
  Baseline-Tibial distal motor latency (ms) | 4.8 (0.6) | 4.9 (0.8) | 4.5 (0.6) | 4.7 (0.7)
  24 Months-Peroneal distal motor latency (ms): number analyzed (Participants) | 26 | 28 | 27 | 28
  24 Months-Peroneal distal motor latency (ms) | 4.3 (0.5) | 4.4 (0.7) | 4.2 (0.7) | 4.2 (0.7)
  24 Months-Sural peak latency (ms): number analyzed (Participants) | 26 | 28 | 27 | 28
  24 Months-Sural peak latency (ms) | 3.5 (0.4) | 3.5 (0.4) | 3.6 (0.6) | 3.4 (0.5)
  24 Months-Tibial distal motor latency (ms): number analyzed (Participants) | 26 | 28 | 27 | 28
  24 Months-Tibial distal motor latency (ms) | 4.3 (0.7) | 4.4 (0.8) | 4.3 (0.9) | 4.6 (1.1)
Statistical Analysis 1: Comparison: Bariatric Surgery/HIIT vs No Bariatric Surgery/Routine Exercise; Measure - Peroneal distal motor latency (ms); Test type: Superiority; p = 0.83, t-test, 2 sided — [p-value comment as in outcome 1, analysis 1]; Mean Difference (Net) = 0.05, 95% CI 2-sided [-0.40 to 0.50]
Statistical Analysis 2: Comparison: Bariatric Surgery/Routine Exercise vs No Bariatric Surgery/Routine Exercise; Measure -Peroneal distal motor latency (ms); Test type: Superiority; p = 0.33, t-test, 2 sided — [p-value comment as in outcome 1, analysis 1]; Mean Difference (Net) = -0.20, 95% CI 2-sided [-0.62 to 0.21]
Statistical Analysis 3: Comparison: No Bariatric Surgery/HIIT vs No Bariatric Surgery/Routine Exercise; Measure -Peroneal distal motor latency (ms); Test type: Superiority; p = 0.75, t-test, 2 sided — [p-value comment as in outcome 1, analysis 1]; Mean Difference (Net) = 0.06, 95% CI 2-sided [-0.36 to 0.49]
Statistical Analysis 4: Comparison: Bariatric Surgery/HIIT vs No Bariatric Surgery/Routine Exercise; Measure - Sural peak latency (ms); Test type: Superiority; p = 0.45, t-test, 2 sided — [p-value comment as in outcome 1, analysis 1]; Mean Difference (Net) = -0.13, 95% CI 2-sided [-0.49 to 0.23]
Statistical Analysis 5: Comparison: Bariatric Surgery/Routine Exercise vs No Bariatric Surgery/Routine Exercise; Measure -Sural peak latency (ms); Test type: Superiority; p = 0.13, t-test, 2 sided — [p-value comment as in outcome 1, analysis 1]; Mean Difference (Net) = -0.24, 95% CI 2-sided [-0.57 to 0.08]
Statistical Analysis 6: Comparison: No Bariatric Surgery/HIIT vs No Bariatric Surgery/Routine Exercise; Measure -Sural peak latency (ms); Test type: Superiority; p = 0.03, t-test, 2 sided — [p-value comment as in outcome 1, analysis 1]; Mean Difference (Net) = -0.41, 95% CI 2-sided [-0.79 to -0.03]
Statistical Analysis 7: Comparison: Bariatric Surgery/HIIT vs No Bariatric Surgery/Routine Exercise; Measure - Tibial distal motor latency (ms); Test type: Superiority; p = 0.05, t-test, 2 sided — [p-value comment as in outcome 1, analysis 1]; Mean Difference (Net) = 0.50, 95% CI 2-sided [-0.002 to 1.01]
Statistical Analysis 8: Comparison: Bariatric Surgery/Routine Exercise vs No Bariatric Surgery/Routine Exercise; Measure - Tibial distal motor latency (ms); Test type: Superiority; p = 0.08, t-test, 2 sided — [p-value comment as in outcome 1, analysis 1]; Mean Difference (Net) = 0.48, 95% CI 2-sided [-0.07 to 1.03]
Statistical Analysis 9: Comparison: No Bariatric Surgery/HIIT vs No Bariatric Surgery/Routine Exercise; Measure - Tibial distal motor latency (ms); Test type: Superiority; p = 0.38, t-test, 2 sided — [p-value comment as in outcome 1, analysis 1]; Mean Difference (Net) = 0.21, 95% CI 2-sided [-0.27 to 0.70]

12. Secondary Outcome: Nerve Conduction Study (NCS) - Motor Amplitude
Description: Amplitude measures the height of electrical signal (waveform) in millivolts produced by the stimulated motor nerve. Was performed on peroneal, and tibial nerves. No response and abnormal values indicate neuropathy.
  * Peroneal: 0 - No response, < 1.1 - Abnormal
  * Tibial: 0 - No response, <1.1 - Abnormal
Time Frame: Baseline and 24 months
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: mV
Arm/Group | Bariatric Surgery/HIIT | Bariatric Surgery/Routine Exercise | No Bariatric Surgery/HIIT | No Bariatric Surgery/Routine Exercise
Number analyzed (Participants) | 35 | 35 | 35 | 35
mV
  Baseline-Peroneal amplitude (mV) | 5.21 (2.39) | 5.95 (3.05) | 5.18 (2.56) | 6.25 (4.13)
  Baseline-Tibial amplitude (mV) | 9.4 (3.59) | 9.16 (4.55) | 8.06 (4.4) | 7.59 (4.66)
  24 Months-Peroneal amplitude (mV): number analyzed (Participants) | 26 | 28 | 27 | 28
  24 Months-Peroneal amplitude (mV) | 4.9 (2.11) | 6.23 (2.93) | 4.93 (2.02) | 5.11 (4.04)
  24 Months-Tibial amplitude (mV): number analyzed (Participants) | 26 | 28 | 27 | 28
  24 Months-Tibial amplitude (mV) | 9.65 (4.98) | 9.28 (4.75) | 8.54 (4.02) | 8.04 (4.22)
Statistical Analysis 1: Comparison: Bariatric Surgery/HIIT vs No Bariatric Surgery/Routine Exercise; Measure - Peroneal amplitude (mV); Test type: Superiority; p = 0.48, t-test, 2 sided — [p-value comment as in outcome 1, analysis 1]
Statistical Analysis 2: Comparison: Bariatric Surgery/Routine Exercise vs No Bariatric Surgery/Routine Exercise; Measure - Peroneal amplitude (mV); Test type: Superiority; p = 0.31, t-test, 2 sided — [p-value comment as in outcome 1, analysis 1]
Statistical Analysis 3: Comparison: No Bariatric Surgery/HIIT vs No Bariatric Surgery/Routine Exercise; Measure - Peroneal amplitude (mV); Test type: Superiority; p = 0.23, t-test, 2 sided — [p-value comment as in outcome 1, analysis 1]
Statistical Analysis 4: Comparison: Bariatric Surgery/HIIT vs No Bariatric Surgery/Routine Exercise; Measure - Tibial amplitude (mV); Test type: Superiority; p = 0.65, t-test, 2 sided — [p-value comment as in outcome 1, analysis 1]
Statistical Analysis 5: Comparison: Bariatric Surgery/Routine Exercise vs No Bariatric Surgery/Routine Exercise; Measure - Tibial amplitude (mV); Test type: Superiority; p = 0.69, t-test, 2 sided — [p-value comment as in outcome 1, analysis 1]
Statistical Analysis 6: Comparison: No Bariatric Surgery/HIIT vs No Bariatric Surgery/Routine Exercise; Measure - Tibial amplitude (mV); Test type: Superiority; p = 0.69, t-test, 2 sided — [p-value comment as in outcome 1, analysis 1]

13. Secondary Outcome: Nerve Conduction Study (NCS) - Sensory Amplitude
Description: Amplitude measures the height of electrical signal (waveform) in microvolts produced by the stimulated sensory nerve. Was performed on sural nerve. No response and abnormal values indicate neuropathy.
  * Sural: 0 - No response, <4 - Abnormal
Time Frame: Baseline and 24 months
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: μV
Arm/Group | Bariatric Surgery/HIIT | Bariatric Surgery/Routine Exercise | No Bariatric Surgery/HIIT | No Bariatric Surgery/Routine Exercise
Number analyzed (Participants) | 35 | 35 | 35 | 35
μV
  Baseline-Sural amplitude (µV) | 12.4 (5) | 10.8 (5.3) | 10.6 (4.7) | 9.1 (5.3)
  24 Months-Sural amplitude (µV): number analyzed (Participants) | 26 | 28 | 27 | 28
  24 Months-Sural amplitude (µV) | 12.4 (6.1) | 14.2 (5.8) | 10.7 (5.7) | 10.6 (6.7)
Statistical Analysis 1: Comparison: Bariatric Surgery/HIIT vs Bariatric Surgery/Routine Exercise; Measure - Sural amplitude (µV); Test type: Superiority; p = 0.82, t-test, 2 sided — [p-value comment as in outcome 1, analysis 1]
Statistical Analysis 2: Comparison: Bariatric Surgery/Routine Exercise vs No Bariatric Surgery/Routine Exercise; Measure - Sural amplitude (µV); Test type: Superiority; p = 0.26, t-test, 2 sided — [p-value comment as in outcome 1, analysis 1]
Statistical Analysis 3: Comparison: No Bariatric Surgery/HIIT vs No Bariatric Surgery/Routine Exercise; Measure - Sural amplitude (µV); Test type: Superiority; p = 0.62, t-test, 2 sided — [p-value comment as in outcome 1, analysis 1]

14. Secondary Outcome: Nerve Conduction Study (NCS) - CV
Description: Conduction velocity (V) measures the speed (m/s) at which the electrical impulse travels along the nerve. Was performed on peroneal nerves. No response and abnormal values indicate neuropathy. Abnormal values are <36 or 39, depending on whether certain criteria applied to the participant. Data was not analyzed separately.
Time Frame: Baseline and 24 months
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: m/s
Arm/Group | Bariatric Surgery/HIIT | Bariatric Surgery/Routine Exercise | No Bariatric Surgery/HIIT | No Bariatric Surgery/Routine Exercise
Number analyzed (Participants) | 35 | 35 | 35 | 35
m/s
  Baseline-Peroneal CV (m/s) | 46.91 (4.14) | 45.37 (4.27) | 46.49 (4.39) | 45.47 (6.38)
  24 Months-Peroneal CV (m/s): number analyzed (Participants) | 26 | 28 | 27 | 28
  24 Months-Peroneal CV (m/s) | 46.96 (5.58) | 47.48 (4.25) | 44.69 (5.43) | 45.96 (5.24)
Statistical Analysis 1: Comparison: Bariatric Surgery/HIIT vs No Bariatric Surgery/Routine Exercise; Measure - Peroneal CV (m/s); Test type: Superiority; p = 0.82, t-test, 2 sided — [p-value comment as in outcome 1, analysis 1]
Statistical Analysis 2: Comparison: Bariatric Surgery/Routine Exercise vs No Bariatric Surgery/Routine Exercise; Measure - Peroneal CV (m/s); Test type: Superiority; p = 0.27, t-test, 2 sided — [p-value comment as in outcome 1, analysis 1]
Statistical Analysis 3: Comparison: No Bariatric Surgery/HIIT vs No Bariatric Surgery/Routine Exercise; Measure - Peroneal CV (m/s); Test type: Superiority; p = 0.52, t-test, 2 sided — [p-value comment as in outcome 1, analysis 1]

15. Secondary Outcome: Nerve Conduction Study (NCS) - F Wave Index
Description: F wave index measures the time in millisecond between stimulation at a distal (near the muscle) point and for the stimulus to travel to the spinal cord and back, allowing to assess the entire length of the nerve.
  Was performed on peroneal, and tibial nerves. No response and abnormal values indicate neuropathy.
  * Peroneal: 0 - No response, >55 - Abnormal
  * Tibial: 0 - No response, >55 - Abnormal
Time Frame: Baseline and 24 months
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: ms
Arm/Group | Bariatric Surgery/HIIT | Bariatric Surgery/Routine Exercise | No Bariatric Surgery/HIIT | No Bariatric Surgery/Routine Exercise
Number analyzed (Participants) | 35 | 35 | 35 | 35
ms
  Baseline-Peroneal F wave index (ms) | 48.29 (6.99) | 49.57 (4.54) | 49.28 (5.73) | 48.91 (9.35)
  Baseline-Tibial F wave index (ms) | 50.84 (8.88) | 51.92 (5.78) | 52.45 (5.4) | 50.8 (9.21)
  24 Months-Peroneal F wave index (ms): number analyzed (Participants) | 26 | 28 | 27 | 28
  24 Months-Peroneal F wave index (ms) | 48.45 (4.57) | 48.5 (5.4) | 48.95 (5.18) | 50.07 (6.95)
  24 Months-Tibial F wave index (ms): number analyzed (Participants) | 26 | 28 | 27 | 28
  24 Months-Tibial F wave index (ms) | 50.56 (5.7) | 50.41 (6.06) | 50.61 (5.32) | 51.88 (5.12)
Statistical Analysis 1: Comparison: Bariatric Surgery/HIIT vs No Bariatric Surgery/Routine Exercise; Measure - Peroneal F wave index (ms); Test type: Superiority; p = 0.32, t-test, 2 sided — [p-value comment as in outcome 1, analysis 1]
Statistical Analysis 2: Comparison: Bariatric Surgery/Routine Exercise vs No Bariatric Surgery/Routine Exercise; Measure - Peroneal F wave index (ms); Test type: Superiority; p = 0.43, t-test, 2 sided — [p-value comment as in outcome 1, analysis 1]
Statistical Analysis 3: Comparison: No Bariatric Surgery/HIIT vs No Bariatric Surgery/Routine Exercise; Measure - Peroneal F wave index (ms); Test type: Superiority; p = 0.48, t-test, 2 sided — [p-value comment as in outcome 1, analysis 1]
Statistical Analysis 4: Comparison: Bariatric Surgery/HIIT vs No Bariatric Surgery/Routine Exercise; Measure - Tibial F wave index (ms); Test type: Superiority; p = 0.75, t-test, 2 sided — [p-value comment as in outcome 1, analysis 1]
Statistical Analysis 5: Comparison: Bariatric Surgery/Routine Exercise vs No Bariatric Surgery/Routine Exercise; Measure - Tibial F wave index (ms); Test type: Superiority; p = 0.09, t-test, 2 sided — [p-value comment as in outcome 1, analysis 1]
Statistical Analysis 6: Comparison: No Bariatric Surgery/HIIT vs No Bariatric Surgery/Routine Exercise; Measure - Tibial F wave index (ms); Test type: Superiority; p = 0.03, t-test, 2 sided — [p-value comment as in outcome 1, analysis 1]

16. Secondary Outcome: Cardiac Autonomic Neuropathy Testing-Deep Breathing/Exhalation to Inhalation (E:I) Ratio
Description: Deep breathing/exhalation to inhalation (E:I) ratio were evaluated using PS monitor software. Values < 1 are abnormal, indicative of cardiovascular autonomic neuropathy
Time Frame: Baseline and 24 months
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: ratio
Arm/Group | Bariatric Surgery/HIIT | Bariatric Surgery/Routine Exercise | No Bariatric Surgery/HIIT | No Bariatric Surgery/Routine Exercise
Number analyzed (Participants) | 35 | 35 | 35 | 35
ratio
  Baseline | 1.3 (0.1) | 1.2 (0.2) | 1.3 (0.2) | 1.2 (0.2)
  24 Months: number analyzed (Participants) | 26 | 28 | 27 | 28
  24 Months | 1.2 (0.2) | 1.3 (0.2) | 1.3 (0.2) | 1.2 (0.2)
Statistical Analysis 1: Comparison: Bariatric Surgery/HIIT vs No Bariatric Surgery/Routine Exercise; Test type: Superiority; p = 0.79, t-test, 2 sided — [p-value comment as in outcome 1, analysis 1]; Mean Difference (Net) = -0.02, 95% CI 2-sided [-0.16 to 0.129]
Statistical Analysis 2: Comparison: Bariatric Surgery/Routine Exercise vs No Bariatric Surgery/Routine Exercise; Test type: Superiority; p = 0.46, t-test, 2 sided — [p-value comment as in outcome 1, analysis 1]; Mean Difference (Net) = -0.05, 95% CI 2-sided [-0.2 to 0.01]
Statistical Analysis 3: Comparison: No Bariatric Surgery/HIIT vs No Bariatric Surgery/Routine Exercise; Test type: Superiority; p = 0.24, t-test, 2 sided — [p-value comment as in outcome 1, analysis 1]; Mean Difference (Net) = -0.01, 95% CI 2-sided [-0.26 to 0.07]
Statistical Analysis 4: Comparison: Bariatric Surgery/HIIT vs No Bariatric Surgery/Routine Exercise; Test type: Superiority; p = 0.98, Mixed Models Analysis — The P-value tests for association between the outcome and treatment at each visit, compared to the no-treatment group; Interaction term for difference in slope = 0.001, 95% CI 2-sided [-0.01 to 0.01]
Statistical Analysis 5: Comparison: Bariatric Surgery/Routine Exercise vs No Bariatric Surgery/Routine Exercise; Test type: Superiority; p = 0.49, Mixed Models Analysis — The P-value tests for association between the outcome and treatment at each visit, compared to the no-treatment group; Interaction term for difference in slope = 0.002, 95% CI 2-sided [-0.004 to 0.01]
Statistical Analysis 6: Comparison: No Bariatric Surgery/HIIT vs No Bariatric Surgery/Routine Exercise; Test type: Superiority; p = 0.17, Mixed Models Analysis — The P-value tests for association between the outcome and treatment at each visit, compared to the no-treatment group; Interaction term for difference in slope = 0.004, 95% CI 2-sided [-0.002 to 0.01]

17. Secondary Outcome: Cardiac Autonomic Neuropathy Testing (30:15 Ratio)
Description: Postural change-30:15 ratio was evaluated using PS monitor software. Values < 1 are abnormal, indicative of cardiovascular autonomic neuropathy
Time Frame: Baseline and 24 months
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: ratio
Arm/Group | Bariatric Surgery/HIIT | Bariatric Surgery/Routine Exercise | No Bariatric Surgery/HIIT | No Bariatric Surgery/Routine Exercise
Number analyzed (Participants) | 35 | 35 | 35 | 35
ratio
  Baseline | 1.1 (0.2) | 1.1 (0) | 1.1 (0.1) | 1.1 (0.1)
  24 Months: number analyzed (Participants) | 26 | 28 | 27 | 28
  24 Months | 1.2 (0.2) | 1.2 (0.2) | 1.2 (0.2) | 1.3 (0.2)
Statistical Analysis 1: Comparison: Bariatric Surgery/HIIT vs No Bariatric Surgery/Routine Exercise; Test type: Superiority; p = 0.07, t-test, 2 sided — [p-value comment as in outcome 1, analysis 1]; Mean Difference (Net) = 0.15, 95% CI 2-sided [-0.01 to 0.31]
Statistical Analysis 2: Comparison: Bariatric Surgery/Routine Exercise vs No Bariatric Surgery/Routine Exercise; Test type: Superiority; p = 0.72, t-test, 2 sided — [p-value comment as in outcome 1, analysis 1]; Mean Difference (Net) = 0.024, 95% CI 2-sided [-0.11 to 0.16]
Statistical Analysis 3: Comparison: No Bariatric Surgery/HIIT vs No Bariatric Surgery/Routine Exercise; Test type: Superiority; p = 0.33, t-test, 2 sided — [p-value comment as in outcome 1, analysis 1]; Mean Difference (Net) = 0.06, 95% CI 2-sided [-0.06 to 0.19]

18. Secondary Outcome: Cardiac Autonomic Neuropathy Testing (Valsalva Ratio)
Description: Valsalva ratio was evaluated using PS monitor software. Values <= 1.10 are abnormal, indicative of cardiovascular autonomic neuropathy
Time Frame: Baseline and 24 months
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: ratio
Arm/Group | Bariatric Surgery/HIIT | Bariatric Surgery/Routine Exercise | No Bariatric Surgery/HIIT | No Bariatric Surgery/Routine Exercise
Number analyzed (Participants) | 35 | 35 | 35 | 35
ratio
  Baseline | 1.5 (0.2) | 1.5 (0.2) | 1.4 (0.2) | 1.4 (0.2)
  24 Months: number analyzed (Participants) | 26 | 28 | 27 | 28
  24 Months | 1.3 (0.2) | 1.4 (0.3) | 1.3 (0.2) | 1.4 (0.3)
Statistical Analysis 1: Comparison: Bariatric Surgery/HIIT vs No Bariatric Surgery/Routine Exercise; Test type: Superiority; p = 0.46, t-test, 2 sided — [p-value comment as in outcome 1, analysis 1]; Mean Difference (Net) = 0.064, 95% CI 2-sided [-0.11 to 0.24]
Statistical Analysis 2: Comparison: Bariatric Surgery/Routine Exercise vs No Bariatric Surgery/Routine Exercise; Test type: Superiority; p = 0.15, t-test, 2 sided — [p-value comment as in outcome 1, analysis 1]; Mean Difference (Net) = 0.13, 95% CI 2-sided [-0.04 to 0.31]
Statistical Analysis 3: Comparison: No Bariatric Surgery/HIIT vs No Bariatric Surgery/Routine Exercise; Test type: Superiority; p = 0.20, t-test, 2 sided — [p-value comment as in outcome 1, analysis 1]; Mean Difference (Net) = 0.11, 95% CI 2-sided [-0.06 to 0.30]

19. Secondary Outcome: Participants With Probable Polyneuropathy as Defined by the Toronto Definition of Probable Neuropathy
Description: Toronto definition of probable neuropathy is having at least 2 out of 3 of the following: abnormal sensory examination, reflexes, and patient-reported symptoms. Data is reported as number of participants who, under the Toronto definition, were identified as having probable polyneuropathy.
Time Frame: 24 months
Population: as for outcome 1
Measure: Number; unit: participants with probable neuropathy
Arm/Group | Bariatric Surgery/HIIT | Bariatric Surgery/Routine Exercise | No Bariatric Surgery/HIIT | No Bariatric Surgery/Routine Exercise
Number analyzed (Participants) | 35 | 35 | 35 | 35
participants with probable neuropathy
  Baseline | 6 | 5 | 9 | 11
  24 Months: number analyzed (Participants) | 26 | 28 | 27 | 28
  24 Months | 9 | 7 | 7 | 9
Statistical Analysis 1: Comparison: Bariatric Surgery/HIIT; Wilcoxon signed rank test was used to compare within-participant change between baseline and 2 year for each treatment group; Test type: Superiority; p = 0.07, Wilcoxon (Mann-Whitney); Wilcoxon test statistic = 10
Statistical Analysis 2: Comparison: Bariatric Surgery/Routine Exercise; [analysis description as in outcome 19, analysis 1]; Test type: Superiority; p = 0.34, Wilcoxon (Mann-Whitney); Wilcoxon test statistic = 3
Statistical Analysis 3: Comparison: No Bariatric Surgery/HIIT; [analysis description as in outcome 19, analysis 1]; Test type: Superiority; p = 0.42, Wilcoxon (Mann-Whitney); Wilcoxon test statistic = 2.5
Statistical Analysis 4: Comparison: No Bariatric Surgery/Routine Exercise; [analysis description as in outcome 19, analysis 1]; Test type: Superiority; p = 0.77, Wilcoxon (Mann-Whitney); Wilcoxon test statistic = 9

20. Secondary Outcome: Michigan Neuropathy Screening Instrument (MNSI)
Description: MNSI questionnaire is scored from 0-15, score > 4 indicate neuropathy, higher scores indicate worse neuropathy.
  A score of 1 point is given for answers of "yes" for questions 1-6, 8-12, 14, and 15 and "no" for questions 7 and 13.
Time Frame: Baseline, 3 month, 12 months and 24 months
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Bariatric Surgery/HIIT | Bariatric Surgery/Routine Exercise | No Bariatric Surgery/HIIT | No Bariatric Surgery/Routine Exercise
Number analyzed (Participants) | 35 | 35 | 35 | 35
score on a scale
  Baseline Questionnaire | 2.5 (2.4) | 2.5 (1.7) | 2.4 (2.2) | 2.8 (2.1)
  3 Months Questionnaire: number analyzed (Participants) | 35 | 32 | 32 | 32
  3 Months Questionnaire | 2.5 (2.7) | 2 (1.9) | 2.5 (2.7) | 2.3 (2.2)
  12 Months Questionnaire: number analyzed (Participants) | 29 | 32 | 28 | 29
  12 Months Questionnaire | 2.7 (2.9) | 2.1 (2.2) | 2.3 (2) | 2.8 (2.1)
  24 Months Questionnaire: number analyzed (Participants) | 26 | 28 | 27 | 28
  24 Months Questionnaire | 3.2 (2.6) | 2.3 (2) | 1.8 (1.7) | 2.8 (2)
Statistical Analysis 1: Comparison: Bariatric Surgery/HIIT vs No Bariatric Surgery/Routine Exercise; Questionnaire; Test type: Superiority; p = 0.21, t-test, 2 sided — [p-value comment as in outcome 1, analysis 1]; Mean Difference (Net) = -0.61, 95% CI 2-sided [-1.5 to 0.35]
Statistical Analysis 2: Comparison: Bariatric Surgery/Routine Exercise vs No Bariatric Surgery/Routine Exercise; Questionnaire; Test type: Superiority; p = 0.85, t-test, 2 sided — [p-value comment as in outcome 1, analysis 1]; Mean Difference (Net) = -0.09, 95% CI 2-sided [-0.98 to 0.80]
Statistical Analysis 3: Comparison: No Bariatric Surgery/HIIT vs No Bariatric Surgery/Routine Exercise; Questionnaire; Test type: Superiority; p = 0.37, t-test, 2 sided — [p-value comment as in outcome 1, analysis 1]; Mean Difference (Net) = 0.46, 95% CI 2-sided [-0.58 to 1.50]
Statistical Analysis 4: Comparison: Bariatric Surgery/HIIT vs No Bariatric Surgery/Routine Exercise; Questionnaire; Test type: Superiority; p = 0.78, Mixed Models Analysis — The P-value tests for association between the outcome and treatment at each visit, compared to the no-treatment group; Interaction term for difference in slope = 1.00, 95% CI 2-sided [0.99 to 1.02]
Statistical Analysis 5: Comparison: Bariatric Surgery/Routine Exercise vs No Bariatric Surgery/Routine Exercise; Questionnaire; Test type: Superiority; p = 0.53, Mixed Models Analysis — The P-value tests for association between the outcome and treatment at each visit, compared to the no-treatment group; Interaction term for difference in slope = 0.99, 95% CI 2-sided [0.98 to 1.01]
Statistical Analysis 6: Comparison: No Bariatric Surgery/HIIT vs No Bariatric Surgery/Routine Exercise; Questionnaire; Test type: Superiority; p = 0.08, Mixed Models Analysis — The P-value tests for association between the outcome and treatment at each visit, compared to the no-treatment group; Interaction term for difference in slope = 0.98, 95% CI 2-sided [0.96 to 1.00]

21. Secondary Outcome: Michigan Neuropathy Screening Instrument (MNSI) - Exam
Description: MNSI exam is scored from 0-8, score >= 2.5 indicate neuropathy. Higher scores indicate worse neuropathy.
Time Frame: Baseline, 3 month, 12 months and 24 months
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Bariatric Surgery/HIIT | Bariatric Surgery/Routine Exercise | No Bariatric Surgery/HIIT | No Bariatric Surgery/Routine Exercise
Number analyzed (Participants) | 35 | 35 | 35 | 35
score on a scale
  Baseline Exam | 1 (1.4) | 0.9 (1.2) | 1.1 (1.4) | 1.3 (1.7)
  3 Months Exam: number analyzed (Participants) | 35 | 32 | 32 | 32
  3 Months Exam | 1 (1.4) | 0.4 (0.7) | 1.2 (1.8) | 1.5 (1.6)
  12 Months Exam: number analyzed (Participants) | 29 | 32 | 28 | 29
  12 Months Exam | 1.1 (1.3) | 1 (1.3) | 1.1 (1.7) | 1.4 (1.7)
  24 Months Exam: number analyzed (Participants) | 26 | 28 | 27 | 28
  24 Months Exam | 0.9 (1.3) | 0.6 (0.9) | 1.3 (1.8) | 1.8 (1.5)
Statistical Analysis 1: Comparison: Bariatric Surgery/HIIT vs No Bariatric Surgery/Routine Exercise; Test type: Superiority; p = 0.01, t-test, 2 sided — [p-value comment as in outcome 1, analysis 1]
Statistical Analysis 2: Comparison: Bariatric Surgery/Routine Exercise vs No Bariatric Surgery/Routine Exercise; Test type: Superiority; p = 0.04, t-test, 2 sided — [p-value comment as in outcome 1, analysis 1]
Statistical Analysis 3: Comparison: No Bariatric Surgery/HIIT vs No Bariatric Surgery/Routine Exercise; Test type: Superiority; p = 0.47, t-test, 2 sided — [p-value comment as in outcome 1, analysis 1]
Statistical Analysis 4: Comparison: Bariatric Surgery/HIIT vs No Bariatric Surgery/Routine Exercise; Test type: Superiority; p = 0.18, Mixed Models Analysis — The P-value tests for association between the outcome and treatment at each visit, compared to the no-treatment group; Interaction term for difference in slope = 0.98, 95% CI 2-sided [0.96 to 1.01]
Statistical Analysis 5: Comparison: Bariatric Surgery/Routine Exercise vs No Bariatric Surgery/Routine Exercise; Test type: Superiority; p = 0.52, Mixed Models Analysis — The P-value tests for association between the outcome and treatment at each visit, compared to the no-treatment group; Interaction term for difference in slope = 0.99, 95% CI 2-sided [0.96 to 1.02]
Statistical Analysis 6: Comparison: No Bariatric Surgery/HIIT vs No Bariatric Surgery/Routine Exercise; Test type: Superiority; p = 0.87, Mixed Models Analysis — The P-value tests for association between the outcome and treatment at each visit, compared to the no-treatment group; Interaction term for difference in slope = 1.00, 95% CI 2-sided [0.97 to 1.02]

22. Secondary Outcome: Michigan Neuropathy Screening Instrument (MNSI) - Index
Description: The Michigan Neuropathy Screening Instrument (MNSI) index is a weighted composite score computed using the sum of the b-coefﬁcients for all items within the MNSI questionnaire (15 questions) and MNSI exam (4 physical/visual exam).
  Range: -0.93, 7.39 Values > 2.5407 are indicative of clinical neuropathy
Time Frame: Baseline, 3 month, 12 months and 24 months
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: MNSI Score
Arm/Group | Bariatric Surgery/HIIT | Bariatric Surgery/Routine Exercise | No Bariatric Surgery/HIIT | No Bariatric Surgery/Routine Exercise
Number analyzed (Participants) | 35 | 35 | 35 | 35
MNSI Score
  Baseline Index | 1.6 (1.3) | 1.5 (0.9) | 1.4 (1.3) | 1.8 (1.3)
  3 Months Index: number analyzed (Participants) | 35 | 32 | 32 | 32
  3 Months Index | 1.6 (1.3) | 1.1 (1) | 1.7 (1.4) | 1.8 (1.5)
  12 Months Index: number analyzed (Participants) | 29 | 32 | 28 | 29
  12 Months Index | 1.7 (1.6) | 1.3 (1.1) | 1.6 (1.3) | 2 (1.5)
  24 Months Index: number analyzed (Participants) | 26 | 28 | 27 | 28
  24 Months Index | 1.7 (1.5) | 1.5 (1.5) | 1.9 (1.3) | 1.9 (1.2)
Statistical Analysis 1: Comparison: Bariatric Surgery/HIIT vs No Bariatric Surgery/Routine Exercise; Test type: Superiority; p = 0.20, t-test, 2 sided — [p-value comment as in outcome 1, analysis 1]
Statistical Analysis 2: Comparison: Bariatric Surgery/Routine Exercise vs No Bariatric Surgery/Routine Exercise; Test type: Superiority; p = 0.57, t-test, 2 sided — [p-value comment as in outcome 1, analysis 1]
Statistical Analysis 3: Comparison: No Bariatric Surgery/HIIT vs No Bariatric Surgery/Routine Exercise; Test type: Superiority; p = 0.61, t-test, 2 sided — [p-value comment as in outcome 1, analysis 1]

23. Secondary Outcome: Utah Early Neuropathy Score (UENS)
Description: UENS is a composite score with five sections measuring multiple clinical measures of nerve injury. Sections are scored separately for each side (Right vs Left), and the total score is the sum across everything. Range: 0-42, higher score represents more severe polyneuropathy.
Time Frame: Baseline, 3 month, 12 months and 24 months
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Bariatric Surgery/HIIT | Bariatric Surgery/Routine Exercise | No Bariatric Surgery/HIIT | No Bariatric Surgery/Routine Exercise
Number analyzed (Participants) | 35 | 35 | 35 | 35
score on a scale
  Baseline UENS Total Score | 2.4 (4.1) | 1.6 (2.6) | 2.4 (3.7) | 3.5 (4.6)
  3 Months UENS Total Score: number analyzed (Participants) | 35 | 32 | 32 | 32
  3 Months UENS Total Score | 1.7 (2.8) | 1.8 (3.5) | 2.9 (5.2) | 3 (4.3)
  12 Months UENS Total Score: number analyzed (Participants) | 29 | 32 | 28 | 29
  12 Months UENS Total Score | 3.9 (4.9) | 2.8 (3.8) | 3.2 (5.2) | 4.8 (6.3)
  24 Months UENS Total Score: number analyzed (Participants) | 26 | 28 | 27 | 28
  24 Months UENS Total Score | 2.8 (3.7) | 2.5 (3.6) | 2.9 (2.3) | 3.8 (4.8)
Statistical Analysis 1: Comparison: Bariatric Surgery/HIIT vs No Bariatric Surgery/Routine Exercise; Total Score; Test type: Superiority; p = 0.44, t-test, 2 sided — [p-value comment as in outcome 1, analysis 1]; Mean Difference (Net) = 0.73, -1.2% CI 2-sided [-1.2 to 2.67]
Statistical Analysis 2: Comparison: Bariatric Surgery/Routine Exercise vs No Bariatric Surgery/Routine Exercise; Total Score; Test type: Superiority; p = 0.97, t-test, 2 sided — [p-value comment as in outcome 1, analysis 1]; Mean Difference (Net) = -0.03, 95% CI 2-sided [-2.16 to 2.10]
Statistical Analysis 3: Comparison: No Bariatric Surgery/HIIT vs No Bariatric Surgery/Routine Exercise; Total Score; Test type: Superiority; p = 0.71, t-test, 2 sided — [p-value comment as in outcome 1, analysis 1]; Mean Difference (Net) = 0.40, 95% CI 2-sided [-1.78 to 2.58]
Statistical Analysis 4: Comparison: Bariatric Surgery/HIIT vs No Bariatric Surgery/Routine Exercise; Total Score; Test type: Superiority; p = 0.99, Mixed Models Analysis — The P-value tests for association between the outcome and treatment at each visit, compared to the no-treatment group; Interaction term for difference in slope = 1.00, 95% CI 2-sided [0.98 to 1.02]
Statistical Analysis 5: Comparison: Bariatric Surgery/Routine Exercise vs No Bariatric Surgery/Routine Exercise; Total Score; Test type: Superiority; p = 0.88, Mixed Models Analysis — The P-value tests for association between the outcome and treatment at each visit, compared to the no-treatment group; Interaction term for difference in slope = 1.00, 95% CI 2-sided [0.98 to 1.02]
Statistical Analysis 6: Comparison: No Bariatric Surgery/HIIT vs No Bariatric Surgery/Routine Exercise; Total Score; Test type: Superiority; p = 0.09, Mixed Models Analysis — The P-value tests for association between the outcome and treatment at each visit, compared to the no-treatment group; Interaction term for difference in slope = 0.99, 95% CI 2-sided [0.97 to 1.00]

24. Secondary Outcome: Modified Toronto Neuropathy Score (mTNS)
Description: mTNS is a scale of 0-33 that measures neuropathy symptoms and exam findings. Higher scores indicate more severe polyneuropathy.
Time Frame: Baseline, 3 month, 12 months and 24 months
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Bariatric Surgery/HIIT | Bariatric Surgery/Routine Exercise | No Bariatric Surgery/HIIT | No Bariatric Surgery/Routine Exercise
Number analyzed (Participants) | 35 | 35 | 35 | 35
score on a scale
  Baseline | 3.8 (7.7) | 1.5 (2.6) | 2.1 (3.4) | 3.5 (5.7)
  3 Months: number analyzed (Participants) | 35 | 32 | 32 | 32
  3 Months | 2.1 (4.2) | 1.3 (1.5) | 2.1 (4.4) | 2.8 (4.7)
  12 Months: number analyzed (Participants) | 29 | 32 | 28 | 29
  12 Months | 3.5 (5.9) | 1.8 (3) | 2.3 (4.1) | 3.4 (5.9)
  24 Months: number analyzed (Participants) | 26 | 28 | 27 | 28
  24 Months | 4.4 (6.4) | 2.6 (2.9) | 1.4 (1.9) | 3.2 (3.9)
Statistical Analysis 1: Comparison: Bariatric Surgery/HIIT vs No Bariatric Surgery/Routine Exercise; Test type: Superiority; p = 0.78, t-test, 2 sided — [p-value comment as in outcome 1, analysis 1]; Mean Difference (Net) = 0.52, 95% CI 2-sided [-3.41 to 4.45]
Statistical Analysis 2: Comparison: Bariatric Surgery/Routine Exercise vs No Bariatric Surgery/Routine Exercise; Test type: Superiority; p = 0.63, t-test, 2 sided — [p-value comment as in outcome 1, analysis 1]; Mean Difference (Net) = -0.59, 95% CI 2-sided [-3.14 to 1.95]
Statistical Analysis 3: Comparison: No Bariatric Surgery/HIIT vs No Bariatric Surgery/Routine Exercise; Test type: Superiority; p = 0.43, t-test, 2 sided — [p-value comment as in outcome 1, analysis 1]; Mean Difference (Net) = 1.01, 95% CI 2-sided [-1.55 to 3.58]
Statistical Analysis 4: Comparison: Bariatric Surgery/HIIT vs No Bariatric Surgery/Routine Exercise; Test type: Superiority; p = 0.43, Mixed Models Analysis — The P-value tests for association between the outcome and treatment at each visit, compared to the no-treatment group; Interaction term for difference in slope = 0.99, 95% CI 2-sided [0.98 to 1.01]
Statistical Analysis 5: Comparison: Bariatric Surgery/Routine Exercise vs No Bariatric Surgery/Routine Exercise; Test type: Superiority; p = 0.83, Mixed Models Analysis — The P-value tests for association between the outcome and treatment at each visit, compared to the no-treatment group; Interaction term for difference in slope = 1.00, 95% CI 2-sided [0.98 to 1.02]
Statistical Analysis 6: Comparison: No Bariatric Surgery/HIIT vs No Bariatric Surgery/Routine Exercise; Test type: Superiority; p < 0.01, Mixed Models Analysis — The P-value tests for association between the outcome and treatment at each visit, compared to the no-treatment group; Interaction term for difference in slope = 0.97, 95% CI 2-sided [0.94 to 0.99]

25. Secondary Outcome: Survey of Autonomic Symptoms (SAS)
Description: SAS evaluates the presence and magnitude of autonomic symptoms. Total impact score ranges from 0-60 (or up to 55 for participants to whom certain criteria did not apply). Higher score indicates worse autonomic neuropathy
Time Frame: Baseline, 3 month, 12 months and 24 months
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Bariatric Surgery/HIIT | Bariatric Surgery/Routine Exercise | No Bariatric Surgery/HIIT | No Bariatric Surgery/Routine Exercise
Number analyzed (Participants) | 35 | 35 | 35 | 35
score on a scale
  Baseline | 4.7 (4.1) | 5 (4.3) | 5.1 (4.7) | 5.1 (5.1)
  3 Months: number analyzed (Participants) | 35 | 32 | 32 | 32
  3 Months | 8.2 (8.3) | 4.9 (4.2) | 3.4 (3.8) | 4.8 (4.3)
  12 Months: number analyzed (Participants) | 29 | 32 | 28 | 29
  12 Months | 5.3 (7.2) | 5.1 (4.1) | 4.5 (3.6) | 6.2 (7.3)
  24 Months: number analyzed (Participants) | 26 | 28 | 27 | 28
  24 Months | 5.3 (7.1) | 8.4 (4) | 5.3 (5.3) | 6.2 (5.7)
Statistical Analysis 1: Comparison: Bariatric Surgery/HIIT vs No Bariatric Surgery/Routine Exercise; Test type: Superiority; p = 0.84, t-test, 2 sided — [p-value comment as in outcome 1, analysis 1]; Mean Difference (Net) = -0.54, 95% CI 2-sided [-6.68 to 5.59]
Statistical Analysis 2: Comparison: Bariatric Surgery/Routine Exercise vs No Bariatric Surgery/Routine Exercise; Test type: Superiority; p = 0.48, t-test, 2 sided — [p-value comment as in outcome 1, analysis 1]; Mean Difference (Net) = 2.70, 95% CI 2-sided [-7.57 to 12.97]
Statistical Analysis 3: Comparison: No Bariatric Surgery/HIIT vs No Bariatric Surgery/Routine Exercise; Test type: Superiority; p = 0.64, t-test, 2 sided — [p-value comment as in outcome 1, analysis 1]; Mean Difference (Net) = -0.87, 95% CI 2-sided [-4.94 to 3.18]

26. Secondary Outcome: Diabetic Neuropathy Score (DNS)
Description: DNS is a questionnaire of neuropathy symptoms. Score ranges 0-4, >/=1 indicates polyneuropathy. 0 indicates no polyneuropathy.
Time Frame: Baseline, 3 month, 12 months and 24 months
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Bariatric Surgery/HIIT | Bariatric Surgery/Routine Exercise | No Bariatric Surgery/HIIT | No Bariatric Surgery/Routine Exercise
Number analyzed (Participants) | 35 | 35 | 35 | 35
score on a scale
  Baseline | 1.1 (1.3) | 0.9 (0.9) | 0.8 (1) | 1.1 (1.4)
  3 Months: number analyzed (Participants) | 35 | 32 | 32 | 32
  3 Months | 1.1 (1.4) | 0.6 (1) | 0.8 (1.2) | 0.9 (1.4)
  12 Moths: number analyzed (Participants) | 29 | 32 | 28 | 29
  12 Moths | 1 (1.3) | 0.6 (0.9) | 0.8 (1.2) | 0.9 (1.1)
  24 Months: number analyzed (Participants) | 26 | 28 | 27 | 28
  24 Months | 1.3 (1.5) | 0.6 (1) | 0.7 (0.8) | 1.1 (1.4)
Statistical Analysis 1: Comparison: Bariatric Surgery/HIIT; Test type: Superiority; p = 0.69, t-test, 2 sided — The P-value tests whether the within-participant change in the group from baseline to 2 years is significant; Mean Difference (Net) = -0.2, Standard Deviation 1.3
Statistical Analysis 2: Comparison: Bariatric Surgery/Routine Exercise; Test type: Superiority; p = 0.24, t-test, 2 sided — The P-value tests whether the within-participant change in the group from baseline to 2 years is significant; Median Difference (Net) = -0.3, Standard Deviation 0.9
Statistical Analysis 3: Comparison: No Bariatric Surgery/HIIT; Test type: Superiority; p = 0.45, t-test, 2 sided — The P-value tests whether the within-participant change in the group from baseline to 2 years is significant; Mean Difference (Net) = -0.2, Standard Deviation 1.1
Statistical Analysis 4: Comparison: No Bariatric Surgery/Routine Exercise; Test type: Superiority; p = 0.84, t-test, 2 sided — The P-value tests whether the within-participant change in the group from baseline to 2 years is significant; Mean Difference (Net) = -0.1, Standard Deviation 1.5

27. Secondary Outcome: Short Form McGill Pain Questionnaire
Description: Sum of the sensory score (0-30) and affective score (0-15) for a total score of 0-45. A higher score represents greater pain present.
Time Frame: Baseline, 3 months, 12 months, 24 months
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Bariatric Surgery/HIIT | Bariatric Surgery/Routine Exercise | No Bariatric Surgery/HIIT | No Bariatric Surgery/Routine Exercise
Number analyzed (Participants) | 35 | 35 | 35 | 35
score on a scale
  Baseline | 3.7 (4.4) | 3.1 (4.4) | 2.7 (4.1) | 3.5 (5.5)
  3 Months: number analyzed (Participants) | 35 | 32 | 32 | 32
  3 Months | 3.8 (7.7) | 2.1 (3.6) | 2.6 (4.2) | 3.5 (6)
  12 Months: number analyzed (Participants) | 29 | 32 | 28 | 29
  12 Months | 3.3 (8.5) | 2.3 (3.4) | 2.4 (2.8) | 2.6 (4.5)
  24 Months: number analyzed (Participants) | 26 | 28 | 27 | 28
  24 Months | 5.2 (6.6) | 2.5 (4.5) | 2.1 (2.6) | 2.2 (3.8)
Statistical Analysis 1: Comparison: Bariatric Surgery/HIIT vs No Bariatric Surgery/Routine Exercise; Mcgill Total Score; Test type: Superiority; p = 0.09, t-test, 2 sided — The P-value tests for association between the outcome and treatment at each visit, compared to the no-treatment group; Mean Difference (Net) = -2.60, 95% CI 2-sided [-5.66 to 0.44]
Statistical Analysis 2: Comparison: Bariatric Surgery/Routine Exercise vs No Bariatric Surgery/Routine Exercise; Mcgill Total Score; Test type: Superiority; p = 0.56, t-test, 2 sided — The P-value tests for association between the outcome and treatment at each visit, compared to the no-treatment group; Mean Difference (Net) = -0.97, 95% CI 2-sided [-4.36 to 2.41]
Statistical Analysis 3: Comparison: No Bariatric Surgery/HIIT vs No Bariatric Surgery/Routine Exercise; Mcgill Total Score; Test type: Superiority; p = 0.21, t-test, 2 sided — The P-value tests for association between the outcome and treatment at each visit, compared to the no-treatment group; Mean Difference (Net) = -1.72, 95% CI 2-sided [-4.5 to 1.05]

28. Secondary Outcome: Numerical Rating Scale for Pain
Description: Participant reported pain scale with range 0-10, higher score indicates more pain.
Time Frame: Baseline, 3 months, 12 months, 24 months
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Bariatric Surgery/HIIT | Bariatric Surgery/Routine Exercise | No Bariatric Surgery/HIIT | No Bariatric Surgery/Routine Exercise
Number analyzed (Participants) | 35 | 35 | 35 | 35
score on a scale
  Baseline | 2.2 (2.6) | 2.7 (3.4) | 2.5 (3.7) | 3.8 (4)
  3 Months: number analyzed (Participants) | 35 | 32 | 32 | 32
  3 Months | 3.3 (4.2) | 2.7 (3.7) | 4.2 (4.2) | 3.6 (4.2)
  12 Months: number analyzed (Participants) | 29 | 32 | 28 | 29
  12 Months | 2.9 (4.0) | 3.5 (4.2) | 6.1 (4.4) | 3.8 (4.4)
  24 Months: number analyzed (Participants) | 26 | 28 | 27 | 28
  24 Months | 3.8 (4.0) | 4.7 (4.7) | 4.5 (4.3) | 5 (4.2)
Statistical Analysis 1: Comparison: Bariatric Surgery/HIIT vs No Bariatric Surgery/Routine Exercise; Test type: Superiority; p = 0.62, t-test, 2 sided — The P-value tests for association between the outcome and treatment at each visit, compared to the no-treatment group
Statistical Analysis 2: Comparison: Bariatric Surgery/Routine Exercise vs No Bariatric Surgery/Routine Exercise; Test type: Superiority; p = 0.92, t-test, 2 sided — The P-value tests for association between the outcome and treatment at each visit, compared to the no-treatment group
Statistical Analysis 3: Comparison: No Bariatric Surgery/HIIT vs No Bariatric Surgery/Routine Exercise; Test type: Superiority; p = 0.90, t-test, 2 sided — The P-value tests for association between the outcome and treatment at each visit, compared to the no-treatment group
Statistical Analysis 4: Comparison: Bariatric Surgery/HIIT vs No Bariatric Surgery/Routine Exercise; Test type: Superiority; p = 0.46, Mixed Models Analysis — The P-value tests for association between the outcome and treatment at each visit, compared to the no-treatment group; Interaction term for difference in slope = -0.02, 95% CI 2-sided [-0.06 to 0.03]
Statistical Analysis 5: Comparison: Bariatric Surgery/Routine Exercise vs No Bariatric Surgery/Routine Exercise; Test type: Superiority; p = 0.47, Mixed Models Analysis — The P-value tests for association between the outcome and treatment at each visit, compared to the no-treatment group; Interaction term for difference in slope = -0.02, 95% CI 2-sided [-0.06 to 0.03]
Statistical Analysis 6: Comparison: No Bariatric Surgery/HIIT vs No Bariatric Surgery/Routine Exercise; Test type: Superiority; p = 0.91, Mixed Models Analysis — The P-value tests for association between the outcome and treatment at each visit, compared to the no-treatment group; Interaction term for difference in slope = 0.003, 95% CI 2-sided [-0.04 to 0.05]

29. Secondary Outcome: Neuropathy Quality of Life (NeuroQOL)
Description: Neuropathy Quality of Life (NeuroQOL) evaluates symptoms and function in regard to quality of life over the past four weeks. Range 1-15, higher score indicates neuropathy having a greater impact on quality of life.
Time Frame: Baseline, 3 months, 12 months, and 24 months
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: NeuroQOL Score
Arm/Group | Bariatric Surgery/HIIT | Bariatric Surgery/Routine Exercise | No Bariatric Surgery/HIIT | No Bariatric Surgery/Routine Exercise
Number analyzed (Participants) | 35 | 35 | 35 | 35
NeuroQOL Score
  Baseline | 2.62 (2.34) | 2.13 (1.12) | 2.1 (0.94) | 2.71 (1.98)
  3 Months: number analyzed (Participants) | 35 | 32 | 32 | 32
  3 Months | 2.49 (2.37) | 1.62 (0.5) | 1.93 (0.97) | 2.7 (1.5)
  12 Months: number analyzed (Participants) | 29 | 32 | 28 | 29
  12 Months | 2.23 (2.48) | 1.62 (0.43) | 2.21 (0.87) | 2.42 (1.26)
  24 Months: number analyzed (Participants) | 26 | 28 | 27 | 28
  24 Months | 3.07 (3.02) | 1.86 (0.86) | 1.7 (0.58) | 2.55 (1.98)
Statistical Analysis 1: Comparison: Bariatric Surgery/HIIT vs No Bariatric Surgery/Routine Exercise; NeuroQOL- overall QOL; Test type: Superiority; p = 0.83, t-test, 2 sided — [p-value comment as in outcome 1, analysis 1]; Mean Difference (Net) = 0.06, 95% CI 2-sided [-0.53 to 0.65]
Statistical Analysis 2: Comparison: Bariatric Surgery/Routine Exercise vs No Bariatric Surgery/Routine Exercise; NeuroQOL- overall QOL; Test type: Superiority; p = 0.97, t-test, 2 sided — [p-value comment as in outcome 1, analysis 1]; Mean Difference (Net) = 0.01, 95% CI 2-sided [-0.76 to 0.78]
Statistical Analysis 3: Comparison: No Bariatric Surgery/HIIT vs No Bariatric Surgery/Routine Exercise; NeuroQOL- overall QOL; Test type: Superiority; p = 0.76, t-test, 2 sided — [p-value comment as in outcome 1, analysis 1]; Mean Difference (Net) = -0.09, 95% CI 2-sided [-0.73 to 0.54]

30. Secondary Outcome: 8 Foot Get Up and Go Test
Description: This test measures in seconds how long it takes the participant to stand up from a seated position, walk around a cone places 8 feet away, and return to the chair and sit down. Less time indicates better speed, agility, and balance when moving.
Time Frame: Baseline, 3 months, 12 months, and 24 months
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: Seconds
Arm/Group | Bariatric Surgery/HIIT | Bariatric Surgery/Routine Exercise | No Bariatric Surgery/HIIT | No Bariatric Surgery/Routine Exercise
Number analyzed (Participants) | 35 | 35 | 35 | 35
Seconds
  Baseline | 6.2 (1.5) | 6.1 (1) | 6.4 (1.2) | 6.6 (1.4)
  3 Months: number analyzed (Participants) | 35 | 32 | 32 | 32
  3 Months | 6 (1.1) | 5.9 (0.8) | 6.4 (1.3) | 6.8 (1.5)
  12 Months: number analyzed (Participants) | 29 | 32 | 28 | 29
  12 Months | 6.2 (1.2) | 5.6 (0.7) | 6.6 (1.6) | 6.8 (1.3)
  24 Months: number analyzed (Participants) | 26 | 28 | 27 | 28
  24 Months | 7.1 (3.9) | 6 (0.9) | 6.5 (1) | 7 (1.2)
Statistical Analysis 1: Comparison: Bariatric Surgery/HIIT; Test type: Superiority; p = 0.58, t-test, 2 sided — The P-value tests whether the within-participant change in the group from baseline to 2 years is significant; Mean Difference (Net) = 0.5, Standard Deviation 2.6
Statistical Analysis 2: Comparison: Bariatric Surgery/Routine Exercise; Test type: Superiority; p = 0.80, t-test, 2 sided — The P-value tests whether the within-participant change in the group from baseline to 2 years is significant; Mean Difference (Net) = -0.1, Standard Deviation 1
Statistical Analysis 3: Comparison: No Bariatric Surgery/HIIT; Test type: Superiority; p = 0.86, t-test, 2 sided — The P-value tests whether the within-participant change in the group from baseline to 2 years is significant; Mean Difference (Net) = 0.1, Standard Deviation 1.4
Statistical Analysis 4: Comparison: No Bariatric Surgery/Routine Exercise; Test type: Superiority; p = 0.46, t-test, 2 sided — The P-value tests whether the within-participant change in the group from baseline to 2 years is significant; Mean Difference (Net) = 0.3, Standard Deviation 1.4

31. Secondary Outcome: Berg Balance Scale
Description: Berg Balance Scale measures participants' ability to balance and avoid falls. Scores range from 0-56, higher score indicates less likely to fall.
Time Frame: Baseline, 3 months, 12 months, and 24 months
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Bariatric Surgery/HIIT | Bariatric Surgery/Routine Exercise | No Bariatric Surgery/HIIT | No Bariatric Surgery/Routine Exercise
Number analyzed (Participants) | 35 | 35 | 35 | 35
score on a scale
  Baseline | 55.41 (1.16) | 55.53 (1.02) | 55.41 (1.16) | 54.57 (1.93)
  3 Months: number analyzed (Participants) | 35 | 32 | 32 | 32
  3 Months | 55.48 (1.5) | 55.47 (1.27) | 55.48 (1.5) | 54.81 (1.73)
  12 Months: number analyzed (Participants) | 29 | 32 | 28 | 29
  12 Months | 54.88 (2.12) | 55.41 (1.48) | 54.88 (2.12) | 54.65 (1.6)
  24 Months: number analyzed (Participants) | 26 | 28 | 27 | 28
  24 Months | 55.15 (2.36) | 55.5 (1.2) | 55.15 (2.36) | 55 (1.89)
Statistical Analysis 1: Comparison: Bariatric Surgery/HIIT; Test type: Superiority; p = 0.38, t-test, 2 sided — The P-value tests whether the within-participant change in the group from baseline to 2 years is significant; Mean Difference (Net) = -0.58, Standard Deviation 2.7
Statistical Analysis 2: Comparison: Bariatric Surgery/Routine Exercise; Test type: Superiority; p = 0.72, t-test, 2 sided — The P-value tests whether the within-participant change in the group from baseline to 2 years is significant; Mean Difference (Net) = 0.11, Standard Deviation 1.15
Statistical Analysis 3: Comparison: No Bariatric Surgery/HIIT; Test type: Superiority; p = 0.55, t-test, 2 sided — The P-value tests whether the within-participant change in the group from baseline to 2 years is significant; Mean Difference (Net) = -0.31, Standard Deviation 2.07
Statistical Analysis 4: Comparison: No Bariatric Surgery/Routine Exercise; Test type: Superiority; p = 0.28, t-test, 2 sided — The P-value tests whether the within-participant change in the group from baseline to 2 years is significant; Mean Difference (Net) = 0.57, Standard Deviation 2.7

32. Secondary Outcome: Modified Falls Efficacy Scale - Fall Evaluation
Description: Patient response indicating if they have fallen in the last year. Data is shown as number of people who have fallen in the last year.
Time Frame: Baseline, 3 months, 12 months, and 24 months
Population: as for outcome 1
Measure: Count of Participants; unit: Participants
Arm/Group | Bariatric Surgery/HIIT | Bariatric Surgery/Routine Exercise | No Bariatric Surgery/HIIT | No Bariatric Surgery/Routine Exercise
Number analyzed (Participants) | 35 | 35 | 35 | 35
Participants
  Baseline | 8 | 9 | 9 | 12
  3 Months: number analyzed (Participants) | 35 | 32 | 32 | 32
  3 Months | 8 | 8 | 8 | 5
  12 Months: number analyzed (Participants) | 29 | 32 | 28 | 29
  12 Months | 7 | 2 | 2 | 10
  24 Months: number analyzed (Participants) | 26 | 28 | 27 | 28
  24 Months | 6 | 8 | 7 | 6
Statistical Analysis 1: Comparison: Bariatric Surgery/HIIT; Test type: Superiority; p = 0.54, t-test, 2 sided — The P-value tests whether the within-participant change in the group from baseline to 2 years is significant
Statistical Analysis 2: Comparison: Bariatric Surgery/Routine Exercise; Test type: Superiority; p = 1.00, t-test, 2 sided — The P-value tests whether the within-participant change in the group from baseline to 2 years is significant
Statistical Analysis 3: Comparison: No Bariatric Surgery/HIIT; Test type: Superiority; p = 0.77, t-test, 2 sided — The P-value tests whether the within-participant change in the group from baseline to 2 years is significant
Statistical Analysis 4: Comparison: No Bariatric Surgery/Routine Exercise; Test type: Superiority; p = 0.24, t-test, 2 sided — The P-value tests whether the within-participant change in the group from baseline to 2 years is significant

33. Secondary Outcome: Neurothesiometer
Description: Neurothesiometer is placed on the bottom of the great toe, and slowly increased until participant reports they can feel the vibration. The greater the microns, the less feeling the participant has, suggestive of worse sensory function.
  Value > 25 Microns is indicative of neuropathy. There is no known maximum range. Lower values indicate better sensory function.
Time Frame: Baseline, 3 months, 12 months, and 24 months
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: Microns
Arm/Group | Bariatric Surgery/HIIT | Bariatric Surgery/Routine Exercise | No Bariatric Surgery/HIIT | No Bariatric Surgery/Routine Exercise
Number analyzed (Participants) | 35 | 35 | 35 | 35
Microns
  Baseline | 8.7 (8.3) | 10.2 (9) | 21.1 (47.4) | 20.2 (34.9)
  3 Months: number analyzed (Participants) | 35 | 32 | 32 | 32
  3 Months | 9.7 (11.3) | 8 (5.6) | 20.8 (47.7) | 15.4 (27)
  12 Months: number analyzed (Participants) | 29 | 32 | 28 | 29
  12 Months | 12.1 (12.8) | 9.9 (15) | 19.1 (47.7) | 23.3 (48.3)
  24 Months: number analyzed (Participants) | 26 | 28 | 27 | 28
  24 Months | 13.6 (14.2) | 8 (6.2) | 12 (11.3) | 21.7 (39.5)
Statistical Analysis 1: Comparison: Bariatric Surgery/HIIT vs No Bariatric Surgery/Routine Exercise; Test type: Superiority; p = 0.36, t-test, 2 sided — [p-value comment as in outcome 1, analysis 1]; Mean Difference (Net) = -2.00, 95% CI 2-sided [-6.37 to 2.36]
Statistical Analysis 2: Comparison: Bariatric Surgery/Routine Exercise vs No Bariatric Surgery/Routine Exercise; Test type: Superiority; p < 0.01, t-test, 2 sided — [p-value comment as in outcome 1, analysis 1]; Mean Difference (Net) = 4.5, 95% CI 2-sided [1.31 to 7.71]
Statistical Analysis 3: Comparison: No Bariatric Surgery/HIIT vs No Bariatric Surgery/Routine Exercise; Test type: Superiority; p = 0.30, t-test, 2 sided — [p-value comment as in outcome 1, analysis 1]; Mean Difference (Net) = 5.62, 95% CI 2-sided [-5.37 to 16.63]

34. Secondary Outcome: NIH Toolbox Cognitive Battery
Description: NIH Toolbox Cognition Fluid (Range: 0-100) - Composite score derived as an average across five cognitive domains.
  It's a fully adjusted T-score comparing the participant to a nationally representative sample, stratified by age and other demographics.
  Individual domain scores are fully adjusted T score with range 0-100 and measures the following-
  * Inhibitory Control and Attention - executive function, attention .
  * Dimensional Change Card Sort - executive function
  * Picture Sequence Memory - episodic memory
  * List Sorting Working Memory - working memory
  * Pattern Comparison - processing speed
  A T-score of 50 represents the population mean. A score of 60 indicates that the participant is 1 SD above the national average for individuals with similar demographic characteristics
  Higher scores reflect better cognitive functionality. No set clinical threshold, scores above mean indicate above average cognition for a given age group.
Time Frame: Baseline and at 24 months
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: T-score
Arm/Group | Bariatric Surgery/HIIT | Bariatric Surgery/Routine Exercise | No Bariatric Surgery/HIIT | No Bariatric Surgery/Routine Exercise
Number analyzed (Participants) | 35 | 35 | 35 | 35
T-score
  Baseline Inhibitory Control and Attention Test | 42.6 (6.8) | 44 (8.3) | 42.7 (7.8) | 43 (8.9)
  Baseline Dimensional Change Card Sort Test | 51.6 (12.9) | 54.6 (11.5) | 54.5 (13.2) | 51.8 (12.3)
  Baseline Picture Sequence Memory Test | 56.2 (11.8) | 55.8 (12.2) | 55.6 (12) | 54.2 (8.5)
  Baseline List Sorting Working Memory Test | 54.8 (10.1) | 51.7 (9.3) | 53.3 (10.8) | 50.3 (8.2)
  Baseline Pattern Comparison Processing Speed Test | 48.9 (13.1) | 49.4 (12.2) | 51 (15) | 50.4 (13.9)
  Baseline Cognition Fluid Composite | 51.2 (12.3) | 51.6 (11.8) | 52.1 (11.2) | 49.8 (11.3)
  24 Months Inhibitory Control and Attention Test: number analyzed (Participants) | 26 | 28 | 27 | 28
  24 Months Inhibitory Control and Attention Test | 42.9 (9.3) | 44.3 (7.6) | 44.2 (8.2) | 43.9 (8.5)
  24 Months Dimensional Change Card Sort Test: number analyzed (Participants) | 26 | 28 | 27 | 28
  24 Months Dimensional Change Card Sort Test | 53.7 (12.5) | 53.7 (13.5) | 56.7 (11) | 54.6 (10.9)
  24 Months Picture Sequence Memory Test: number analyzed (Participants) | 26 | 28 | 27 | 28
  24 Months Picture Sequence Memory Test | 55.9 (10.8) | 54.7 (13) | 58.7 (10.8) | 56.3 (10.8)
  24 Months List Sorting Working Memory Test: number analyzed (Participants) | 26 | 28 | 27 | 28
  24 Months List Sorting Working Memory Test | 56.6 (10.1) | 52.1 (8.6) | 54.4 (7.5) | 50.7 (11.4)
  24 Months Pattern Comparison Processing Speed Test: number analyzed (Participants) | 26 | 28 | 27 | 28
  24 Months Pattern Comparison Processing Speed Test | 52.7 (13.8) | 46.7 (16.7) | 48.8 (13.4) | 47.3 (15.7)
  24 Months Cognition Fluid Composite: number analyzed (Participants) | 26 | 28 | 27 | 28
  24 Months Cognition Fluid Composite | 53.5 (12.2) | 50.4 (11.2) | 53.9 (9.1) | 50.6 (10.2)
Statistical Analysis 1: Comparison: Bariatric Surgery/HIIT vs No Bariatric Surgery/Routine Exercise; Inhibitory Control and Attention Test; Test type: Superiority; p = 0.16, t-test, 2 sided — [p-value comment as in outcome 1, analysis 1]; Mean Difference (Net) = 3.14, 95% CI 2-sided [-1.30 to 7.58]
Statistical Analysis 2: Comparison: Bariatric Surgery/Routine Exercise vs No Bariatric Surgery/Routine Exercise; Inhibitory Control and Attention Test; Test type: Superiority; p = 0.33, t-test, 2 sided — [p-value comment as in outcome 1, analysis 1]; Mean Difference (Net) = 1.91, 95% CI 2-sided [-2.05 to 5.88]
Statistical Analysis 3: Comparison: No Bariatric Surgery/HIIT vs No Bariatric Surgery/Routine Exercise; Inhibitory Control and Attention Test; Test type: Superiority; p = 0.49, t-test, 2 sided — [p-value comment as in outcome 1, analysis 1]; Mean Difference (Net) = 1.43, 95% CI 2-sided [-2.72 to 5.59]
Statistical Analysis 4: Comparison: Bariatric Surgery/HIIT vs No Bariatric Surgery/Routine Exercise; Dimensional Change Card Sort Test; Test type: Superiority; p = 0.35, t-test, 2 sided — [p-value comment as in outcome 1, analysis 1]; Mean Difference (Net) = 2.97, 95% CI 2-sided [-3.48 to 9.44]
Statistical Analysis 5: Comparison: Bariatric Surgery/Routine Exercise vs No Bariatric Surgery/Routine Exercise; Dimensional Change Card Sort Test; Test type: Superiority; p = 0.10, t-test, 2 sided — [p-value comment as in outcome 1, analysis 1]; Mean Difference (Net) = 5.6, 95% CI 2-sided [-3.48 to 9.44]
Statistical Analysis 6: Comparison: No Bariatric Surgery/HIIT vs No Bariatric Surgery/Routine Exercise; Dimensional Change Card Sort Test; Test type: Superiority; p = 0.32, t-test, 2 sided — [p-value comment as in outcome 1, analysis 1]; Mean Difference (Net) = 3.24, 95% CI 2-sided [-3.34 to 9.82]
Statistical Analysis 7: Comparison: Bariatric Surgery/HIIT vs No Bariatric Surgery/Routine Exercise; Picture Sequence Memory Test; Test type: Superiority; p = 0.49, t-test, 2 sided — [p-value comment as in outcome 1, analysis 1]; Mean Difference (Net) = 2.4, 95% CI 2-sided [-4.57 to 9.37]
Statistical Analysis 8: Comparison: Bariatric Surgery/Routine Exercise vs No Bariatric Surgery/Routine Exercise; Picture Sequence Memory Test; Test type: Superiority; p = 0.30, t-test, 2 sided — [p-value comment as in outcome 1, analysis 1]; Mean Difference (Net) = 3.2, 95% CI 2-sided [-3.03 to 9.56]
Statistical Analysis 9: Comparison: No Bariatric Surgery/HIIT vs No Bariatric Surgery/Routine Exercise; Picture Sequence Memory Test; Test type: Superiority; p = 0.86, t-test, 2 sided — [p-value comment as in outcome 1, analysis 1]; Median Difference (Net) = 0.49, 95% CI 2-sided [-5.40 to 6.38]
Statistical Analysis 10: Comparison: Bariatric Surgery/HIIT vs No Bariatric Surgery/Routine Exercise; List Sorting Working Memory Test; Test type: Superiority; p = 0.88, t-test, 2 sided — [p-value comment as in outcome 1, analysis 1]; Mean Difference (Net) = 0.42, 95% CI 2-sided [-5.39 to 6.24]
Statistical Analysis 11: Comparison: Bariatric Surgery/Routine Exercise vs No Bariatric Surgery/Routine Exercise; List Sorting Working Memory Test; Test type: Superiority; p = 0.83, t-test, 2 sided — [p-value comment as in outcome 1, analysis 1]; Mean Difference (Net) = 0.60, 95% CI 2-sided [-5.14 to 6.31]
Statistical Analysis 12: Comparison: No Bariatric Surgery/HIIT vs No Bariatric Surgery/Routine Exercise; List Sorting Working Memory Test; Test type: Superiority; p = 0.81, t-test, 2 sided — [p-value comment as in outcome 1, analysis 1]; Mean Difference (Net) = -0.62, 95% CI 2-sided [-6.02 to 4.76]
Statistical Analysis 13: Comparison: Bariatric Surgery/HIIT vs No Bariatric Surgery/Routine Exercise; Pattern Comparison Processing Speed Test; Test type: Superiority; p = 0.12, t-test, 2 sided — [p-value comment as in outcome 1, analysis 1]; Mean Difference (Net) = -5.29, 95% CI 2-sided [-12.1 to 1.57]
Statistical Analysis 14: Comparison: Bariatric Surgery/Routine Exercise vs No Bariatric Surgery/Routine Exercise; Pattern Comparison Processing Speed Test; Test type: Superiority; p = 0.63, t-test, 2 sided — [p-value comment as in outcome 1, analysis 1]; Mean Difference (Net) = -1.84, 95% CI 2-sided [-9.53 to 5.84]
Statistical Analysis 15: Comparison: No Bariatric Surgery/HIIT vs No Bariatric Surgery/Routine Exercise; Pattern Comparison Processing Speed Test; Test type: Superiority; p = 0.40, t-test, 2 sided — [p-value comment as in outcome 1, analysis 1]; Mean Difference (Net) = -2.87, 95% CI 2-sided [-9.80 to 4.05]
Statistical Analysis 16: Comparison: Bariatric Surgery/HIIT vs No Bariatric Surgery/Routine Exercise; Cognition Fluid Composite; Test type: Superiority; p = 0.65, t-test, 2 sided — [p-value comment as in outcome 1, analysis 1]; Mean Difference (Net) = 1.04, 95% CI 2-sided [-3.63 to 5.73]
Statistical Analysis 17: Comparison: Bariatric Surgery/Routine Exercise vs No Bariatric Surgery/Routine Exercise; Cognition Fluid Composite; Test type: Superiority; p = 0.27, t-test, 2 sided — [p-value comment as in outcome 1, analysis 1]; Mean Difference (Net) = 2.68, 95% CI 2-sided [-2.17 to 7.54]
Statistical Analysis 18: Comparison: No Bariatric Surgery/HIIT vs No Bariatric Surgery/Routine Exercise; Cognition Fluid Composite; Test type: Superiority; p = 0.90, t-test, 2 sided — [p-value comment as in outcome 1, analysis 1]; Mean Difference (Net) = 0.27, 95% CI 2-sided [-4.10 to 4.65]
Statistical Analysis 19: Comparison: Bariatric Surgery/HIIT vs No Bariatric Surgery/Routine Exercise; Cognition Fluid Composite; Test type: Superiority; p = 0.85, Mixed Models Analysis — The P-value tests for association between the outcome and treatment at each visit, compared to the no-treatment group; Interaction term for difference in slope = -0.02, 95% CI 2-sided [-0.21 to 0.17]
Statistical Analysis 20: Comparison: Bariatric Surgery/Routine Exercise vs No Bariatric Surgery/Routine Exercise; Cognition Fluid Composite; Test type: Superiority; p = 0.28, Mixed Models Analysis — The P-value tests for association between the outcome and treatment at each visit, compared to the no-treatment group; Interaction term for difference in slope = -0.10, 95% CI 2-sided [-0.29 to 0.09]
Statistical Analysis 21: Comparison: No Bariatric Surgery/HIIT vs No Bariatric Surgery/Routine Exercise; Cognition Fluid Composite; Test type: Superiority; p = 0.99, Mixed Models Analysis — The P-value tests for association between the outcome and treatment at each visit, compared to the no-treatment group; Mean Difference (Net) = 0.001, 95% CI 2-sided [-0.18 to 0.19]

35. Secondary Outcome: Rey Auditory Verbal Learning Test
Description: Used to evaluate verbal learning and memory using a list of 15 unrelated words presented to the participant over repeat trial.
  Includes 3 independent scales:
  * Auditory Learning (Total recall) - Measures memory and learning ability. Raw score range (0- 75)
  * Delayed Recall - Measures long term memory retention. Raw score range (0-15)
  * Recognition - Measures ability to recognize previously learned information. Raw score range (0-15).
  * Raw scores were converted to age-standardized Z-scores using 10-year age bands (e.g., 20-29, 30-39, 40-49, etc.), with a mean of 0 and standard deviation of 1.
  * A Z-score of 0 represents the population mean
  * For each scale, scores above 0 are better. Standard deviations above the mean indicates a better learning and memory ability for a given age group.
  No set clinical threshold, scores above mean indicate above average cognition for a given age group.
Time Frame: Baseline and at 24 months
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: Z-score
Arm/Group | Bariatric Surgery/HIIT | Bariatric Surgery/Routine Exercise | No Bariatric Surgery/HIIT | No Bariatric Surgery/Routine Exercise
Number analyzed (Participants) | 35 | 35 | 35 | 35
Z-score
  Baseline Auditory Learning | 0.1 (1.2) | 0.3 (1.2) | 0.4 (0.8) | 0.4 (1)
  Baseline Delayed Recall | 0 (1.1) | -0.2 (1.1) | 0.1 (0.9) | -0.1 (1)
  Baseline Recognition | 0.7 (0.8) | 0.6 (0.8) | 0.7 (1.2) | 0.7 (0.9)
  24 Months Auditory Learning: number analyzed (Participants) | 26 | 28 | 27 | 27
  24 Months Auditory Learning | -0.2 (1.3) | 0.2 (1.2) | 0.4 (1) | 0 (1.1)
  24 Months Delayed Recall: number analyzed (Participants) | 26 | 28 | 27 | 27
  24 Months Delayed Recall | -0.4 (1) | -0.1 (1) | 0.2 (0.9) | -0.1 (1.1)
  24 Months Recognition: number analyzed (Participants) | 26 | 28 | 27 | 27
  24 Months Recognition | 0.6 (1.2) | 0.9 (0.8) | 0.8 (1.2) | 0 (1)
Statistical Analysis 1: Comparison: Bariatric Surgery/HIIT vs No Bariatric Surgery/Routine Exercise; Auditory Learning; Test type: Superiority; p = 0.57, t-test, 2 sided — [p-value comment as in outcome 1, analysis 1]; Mean Difference (Net) = -0.19, 95% CI 2-sided [-0.87 to 0.49]
Statistical Analysis 2: Comparison: Bariatric Surgery/Routine Exercise vs No Bariatric Surgery/Routine Exercise; Auditory Learning; Test type: Superiority; p = 0.33, t-test, 2 sided — [p-value comment as in outcome 1, analysis 1]; Mean Difference (Net) = -0.26, 95% CI 2-sided [-0.81 to 0.28]
Statistical Analysis 3: Comparison: No Bariatric Surgery/HIIT vs No Bariatric Surgery/Routine Exercise; Auditory Learning; Test type: Superiority; p = 0.22, t-test, 2 sided — [p-value comment as in outcome 1, analysis 1]; Median Difference (Net) = -0.38, 95% CI 2-sided [-1.00 to 0.23]
Statistical Analysis 4: Comparison: Bariatric Surgery/HIIT vs No Bariatric Surgery/Routine Exercise; Delayed Recall; Test type: Superiority; p = 0.27, t-test, 2 sided — [p-value comment as in outcome 1, analysis 1]; Mean Difference (Net) = 0.29, 95% CI 2-sided [-0.23 to 0.81]
Statistical Analysis 5: Comparison: Bariatric Surgery/Routine Exercise vs No Bariatric Surgery/Routine Exercise; Delayed Recall; Test type: Superiority; p = 0.54, t-test, 2 sided — [p-value comment as in outcome 1, analysis 1]; Mean Difference (Net) = -0.16, 95% CI 2-sided [-0.69 to 0.37]
Statistical Analysis 6: Comparison: No Bariatric Surgery/HIIT vs No Bariatric Surgery/Routine Exercise; Delayed Recall; Test type: Superiority; p = 0.93, t-test, 2 sided — [p-value comment as in outcome 1, analysis 1]; Mean Difference (Net) = -0.02, 95% CI 2-sided [-0.57 to 0.53]
Statistical Analysis 7: Comparison: Bariatric Surgery/HIIT vs No Bariatric Surgery/Routine Exercise; Recognition; Test type: Superiority; p = 0.64, t-test, 2 sided — [p-value comment as in outcome 1, analysis 1]; Mean Difference (Net) = 0.14, 95% CI 2-sided [-0.46 to 0.74]
Statistical Analysis 8: Comparison: Bariatric Surgery/Routine Exercise vs No Bariatric Surgery/Routine Exercise; Recognition; Test type: Superiority; p = 0.37, t-test, 2 sided — [p-value comment as in outcome 1, analysis 1]; Mean Difference (Net) = -0.21, 95% CI 2-sided [-0.70 to 0.27]
Statistical Analysis 9: Comparison: No Bariatric Surgery/HIIT vs No Bariatric Surgery/Routine Exercise; Recognition; Test type: Superiority; p = 0.88, t-test, 2 sided — [p-value comment as in outcome 1, analysis 1]; Mean Difference (Net) = 0.04, 95% CI 2-sided [-0.59 to 0.69]

ADVERSE EVENTS:
Time Frame: 2 years
Description: Participants who withdrew from the study were not tracked after their withdrawal date
Arm/Group | Bariatric Surgery/HIIT | No Bariatric Surgery/HIIT | Bariatric Surgery/Routine Exercise | No Bariatric Surgery/Routine Exercise
All-Cause Mortality (participants affected / at risk) | 0/35 | 0/35 | 0/35 | 0/35
Serious Adverse Events (participants affected / at risk) | 0/35 | 0/35 | 0/35 | 0/35
Other Adverse Events (participants affected / at risk) | 0/35 | 2/35 | 1/35 | 0/35
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Bariatric Surgery/HIIT (N=35) | No Bariatric Surgery/HIIT (N=35) | Bariatric Surgery/Routine Exercise (N=35) | No Bariatric Surgery/Routine Exercise (N=35)
Infection at Skin Biopsy Site (Infections and infestations) | 0 (0) | 1 (1) | 1 (1) | 0 (0)
Injury During Exercise (Injury, poisoning and procedural complications) | 0 (0) | 1 (1) | 0 (0) | 0 (0)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (3):
  • Study Protocol (2020-07-08): https://cdn.clinicaltrials.gov/large-docs/85/NCT03617185/Prot_000.pdf
  • Statistical Analysis Plan (2025-07-02): https://cdn.clinicaltrials.gov/large-docs/85/NCT03617185/SAP_001.pdf
  • Informed Consent Form (2024-02-22): https://cdn.clinicaltrials.gov/large-docs/85/NCT03617185/ICF_002.pdf